CLINICAL TRIAL: NCT02885246
Title: Prevalence, Strain Circulation and Disease Burden of Seasonal Influenza A and B in Panama, Selected Countries of Central America and the Caribbean From the Year 2010 to 2015
Brief Title: Prevalence, Strain Circulation and Disease Burden Study of Seasonal Influenza A and B in Panama, Selected Countries of Central America and the Caribbean From the Year 2010 to 2015
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 205049
Record Dates: First submitted 2016-08-26; First posted 2016-08-31 (Estimated); Results first posted 2020-03-03 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-03

CONDITIONS: Influenza, Human
Keywords: Panama; Influenza B; Influenza A; Strain circulation; Database
MeSH Terms: conditions — Influenza, Human | interventions — Data Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Influenza Virus Positive Group: The group included specimen samples with a laboratory confirmed diagnosis of influenza A and/or B, reported in the Instituto Conmemorativo Gorgas de Estudios de la Salud (ICGES) database of Panama, from January 2011 to December 2017.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — The ICGES database of Panama will be checked for all seasonal influenza A and/or B positive cases reported via influenza surveillance programs from 2010 to 2015.

SUMMARY:
The purpose of this study is to assess the prevalence, strain circulation and disease burden of seasonal Influenza A and B in Panama, selected countries of Central America and the Caribbean from the Year 2010 to 2015.

DETAILED DESCRIPTION:
The Gorgas Memorial Institute for Health Studies (ICGES) is a public health institution established in Panama dedicated to health research and disease prevention. It has been performing virological isolations of influenza and is a part of the World Health Organisation (WHO) Global Influenza Surveillance and Response System (GISRS) and a direct collaborator of the Centre for Disease Control and Prevention (CDC).

From 2010 a sentinel surveillance program is being conducted in Panama within the ICGES to collect data on influenza and other respiratory viruses using CDC guidance for Respiratory Disease Surveillance. This study aims to utilize this data source for analyzing the burden of influenza within the region.

ELIGIBILITY:
Inclusion Criteria:

* All subjects diagnosed with seasonal influenza A and/or B, reported in the ICGES database of Panama, from January 2010 to December 2015.

Exclusion Criteria:

* N/A.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The Total population will include all subjects included in the study. Information will only be collected for all eligible subjects (aggregated) captured by the ICGES Database.
Sampling Method: Non-Probability Sample
Enrollment: 1839 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2018-09-17 (Actual); Study Completion 2018-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Panama City, Panama

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a database study with no subject enrollment. The seasonal influenza A and/or B cases reported in the study centers were recorded in country specific national influenza surveillance program databases. Data were not available for selected countries of Central America and the Caribbean. Therefore,only data from Panama were analysed.
Pre-assignment Details: All data was taken from the Instituto Conmemorativo Gorgas de Estudios de la Salud (ICGES) database of Panama, from January 2011 to December 2017. Based on the dates of data transfer and data availability, the data collection period was updated as January 2011-December 2017 instead of January 2010-December 2015, previously defined per protocol.
Period: Overall Study
Arm/Group | Influenza Virus Positive Group
Started | 1839
Completed | 1839
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Influenza Virus Positive Group
Number analyzed (Participants) | 1839
Age, Customized [Count of Participants; unit: Participants]
  <2 years | 567
  2-4 years | 170
  5-19 years | 283
  20-39 years | 313
  40-59 years | 291
  ≥60 years | 190
  Unspecified | 25
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 905
  Female | 909
  Unspecified | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Seasonal Influenza A and /or B Cases by Age Group, in Panama (Using the Data Reported Via National Influenza Surveillance Program)
Description: The case definition of Influenza was any clinical specimen confirmed by a positive laboratory test. Cases were stratified by the following age categories: less than (<) 2 years; 2-4 years; 5-19 years; 20-39 years; 40-59 years; greater than of equal to (≥) 60 years and Unspecified age, instead of <1, 1-4, 5-9, 10-14, 15-19, 20-24, 25-44, 45-49, 50-59, 60-64 and ≥ 65 years, as initially described in the Protocol. Note that one specimen sample was positive for both influenza A and B so the number started still remains 1839.
Time Frame: From January 2011 to December 2017
Population: The analysis was performed on the Total Cohort which included all specimen samples diagnosed with seasonal influenza A and/or B, reported in the ICGES database of Panama, from January 2011 to December 2017.
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza Virus Positive Group
Number analyzed (Participants) | 1839
Participants
  Influenza A <2 years: number analyzed (Participants) | 567
  Influenza A <2 years | 448
  Influenza B <2 years: number analyzed (Participants) | 567
  Influenza B <2 years | 120
  Influenza A 2-4 years: number analyzed (Participants) | 170
  Influenza A 2-4 years | 123
  Influenza B 2-4 years: number analyzed (Participants) | 170
  Influenza B 2-4 years | 47
  Influenza A 5-19 years: number analyzed (Participants) | 283
  Influenza A 5-19 years | 170
  Influenza B 5-19 years: number analyzed (Participants) | 283
  Influenza B 5-19 years | 113
  Influenza A 20-39 years: number analyzed (Participants) | 313
  Influenza A 20-39 years | 274
  Influenza B 20-39 years: number analyzed (Participants) | 313
  Influenza B 20-39 years | 39
  Influenza A 40-59 years: number analyzed (Participants) | 291
  Influenza A 40-59 years | 254
  Influenza B 40-59 years: number analyzed (Participants) | 291
  Influenza B 40-59 years | 37
  Influenza A ≥60: number analyzed (Participants) | 190
  Influenza A ≥60 | 180
  Influenza B ≥60: number analyzed (Participants) | 190
  Influenza B ≥60 | 10
  Influenza A Unspecified: number analyzed (Participants) | 25
  Influenza A Unspecified | 15
  Influenza B Unspecified: number analyzed (Participants) | 25
  Influenza B Unspecified | 10
  Influenza A Total | 1464
  Influenza B Total | 376

2. Primary Outcome: Number of Seasonal Influenza A Cases by Virus Subtypes, in Panama (Using the Data Reported Via National Influenza Surveillance Program) Among All Influenza Cases A and/or B
Description: The case definition of Influenza was any clinical specimen confirmed by a positive laboratory test. Cases were stratified by virus subtype (H1N1 and H3N2) and the following age categories: less than (<) 2 years; 2-4 years; 5-19 years; 20-39 years; 40-59 years; greater than of equal to (≥) 60 years. Note that one specimen sample was positive for both influenza A and B so the number started still remains 1839.
Time Frame: From January 2011 to December 2017
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza Virus Positive Group
Number analyzed (Participants) | 1839
Participants
  H1N1 <2 years: number analyzed (Participants) | 567
  H1N1 <2 years | 259
  H3N2 <2 years: number analyzed (Participants) | 567
  H3N2 <2 years | 189
  H1N1 2-4 years: number analyzed (Participants) | 170
  H1N1 2-4 years | 80
  H3N2 2-4 years: number analyzed (Participants) | 170
  H3N2 2-4 years | 43
  H1N1 5-19 years: number analyzed (Participants) | 283
  H1N1 5-19 years | 119
  H3N2 5-19 years: number analyzed (Participants) | 283
  H3N2 5-19 years | 51
  H1N1 20-39 years: number analyzed (Participants) | 313
  H1N1 20-39 years | 199
  H3N2 20-39 years: number analyzed (Participants) | 313
  H3N2 20-39 years | 75
  H1N1 40-59 years: number analyzed (Participants) | 291
  H1N1 40-59 years | 201
  H3N2 40-59 years: number analyzed (Participants) | 291
  H3N2 40-59 years | 53
  H1N1 ≥60 years: number analyzed (Participants) | 190
  H1N1 ≥60 years | 137
  H3N2 ≥60 years: number analyzed (Participants) | 190
  H3N2 ≥60 years | 43
  H1N1 Unspecified: number analyzed (Participants) | 25
  H1N1 Unspecified | 12
  H3N2 Unspecified: number analyzed (Participants) | 25
  H3N2 Unspecified | 3
  H1N1 Total | 1007
  H3N2 Total | 457

3. Primary Outcome: Number of Seasonal Influenza B Cases by Strain Lineage, in Panama (Using the Data Reported Via National Influenza Surveillance Program) Among All Influenza Cases A and/or B
Description: The case definition of Influenza was any clinical specimen confirmed by a positive laboratory test. Cases were stratified by lineage (Victoria and Yamagata) and the following age categories: less than (<) 2 years; 2-4 years; 5-19 years; 20-39 years; 40-59 years; greater than of equal to (≥) 60 years. Note that one specimen sample was positive for both influenza A and B so the number started still remains 1839.
Time Frame: From January 2011 to December 2017
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza Virus Positive Group
Number analyzed (Participants) | 1839
Participants
  Victoria < 2 years: number analyzed (Participants) | 567
  Victoria < 2 years | 90
  Yamagata < 2 years: number analyzed (Participants) | 567
  Yamagata < 2 years | 30
  Victoria 2-4 years: number analyzed (Participants) | 170
  Victoria 2-4 years | 36
  Yamagata 2-4 years: number analyzed (Participants) | 170
  Yamagata 2-4 years | 11
  Victoria 5-19 years: number analyzed (Participants) | 283
  Victoria 5-19 years | 84
  Yamagata 5-19 years: number analyzed (Participants) | 283
  Yamagata 5-19 years | 29
  Victoria 20-39 years: number analyzed (Participants) | 313
  Victoria 20-39 years | 30
  Yamagata 20-39 years: number analyzed (Participants) | 313
  Yamagata 20-39 years | 9
  Victoria 40-59 years: number analyzed (Participants) | 291
  Victoria 40-59 years | 13
  Yamagata 40-59 years: number analyzed (Participants) | 291
  Yamagata 40-59 years | 24
  Victoria ≥60 years: number analyzed (Participants) | 190
  Victoria ≥60 years | 8
  Yamagata ≥60 years: number analyzed (Participants) | 190
  Yamagata ≥60 years | 2
  Victoria Unspecified: number analyzed (Participants) | 25
  Victoria Unspecified | 8
  Yamagata Unspecified: number analyzed (Participants) | 25
  Yamagata Unspecified | 2
  Victoria Total | 269
  Yamagata Total | 107

4. Secondary Outcome: Number of Cases With Laboratory Confirmed Diagnosis Seasonal Influenza A and/or B Who Experienced Clinical Features (Clinical Symptoms)
Description: The signs and symptoms assessed were: Fever, Cough, Sore throat, Rhinorrhea, Dyspnea, Vomiting, Diarrhea, Myalgias, Nausea, Headache, Wheezing, Apnea, Tachypnea, Polypnea, Arthralgia, Chest Pain, Convulsion, Hyporexia, Weakness, Irritability, Odynophagia, Abdominal pain, Conjunctivitis, Cyanosis and Chills. Each sign and symptom was assessed in four categories: yes = presence of sign/symptom; no = absence of sign/symptom; form not filled = no epi surveillance form available; and unspecified= no data on the Epi surveillance form. Analysis related to duration of the illness was not performed as the data was not collected. Note that one specimen sample was positive for both influenza A and B so the number started still remains 1839.
Time Frame: From January 2011 to December 2017
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza Virus Positive Group
Number analyzed (Participants) | 1839
Participants
  Fever-Yes (2011): number analyzed (Participants) | 47
  Fever-Yes (2011) | 41
  Fever-No (2011): number analyzed (Participants) | 47
  Fever-No (2011) | 4
  Fever-Form not filled (2011): number analyzed (Participants) | 47
  Fever-Form not filled (2011) | 0
  Fever-Unspecified (2011): number analyzed (Participants) | 47
  Fever-Unspecified (2011) | 2
  Cough-Yes (2011): number analyzed (Participants) | 47
  Cough-Yes (2011) | 40
  Cough-No (2011): number analyzed (Participants) | 47
  Cough-No (2011) | 4
  Cough-Form not filled (2011): number analyzed (Participants) | 47
  Cough-Form not filled (2011) | 0
  Cough-Unspecified (2011): number analyzed (Participants) | 47
  Cough-Unspecified (2011) | 3
  Sore throat-Yes (2011): number analyzed (Participants) | 47
  Sore throat-Yes (2011) | 26
  Sore throat-No (2011): number analyzed (Participants) | 47
  Sore throat-No (2011) | 18
  Sore throat-Form not filled (2011): number analyzed (Participants) | 47
  Sore throat-Form not filled (2011) | 0
  Sore throat-Unspecified (2011): number analyzed (Participants) | 47
  Sore throat-Unspecified (2011) | 3
  Rhinorrhea-Yes (2011): number analyzed (Participants) | 47
  Rhinorrhea-Yes (2011) | 41
  Rhinorrhea-No (2011): number analyzed (Participants) | 47
  Rhinorrhea-No (2011) | 3
  Rhinorrhea-Form not filled (2011): number analyzed (Participants) | 47
  Rhinorrhea-Form not filled (2011) | 0
  Rhinorrhea-Unspecified (2011): number analyzed (Participants) | 47
  Rhinorrhea-Unspecified (2011) | 3
  Dyspnea-Yes (2011): number analyzed (Participants) | 47
  Dyspnea-Yes (2011) | 4
  Dyspnea-No (2011): number analyzed (Participants) | 47
  Dyspnea-No (2011) | 32
  Dyspnea-Form not filled (2011): number analyzed (Participants) | 47
  Dyspnea-Form not filled (2011) | 0
  Dyspnea-Unspecified (2011): number analyzed (Participants) | 47
  Dyspnea-Unspecified (2011) | 11
  Vomiting-Yes (2011): number analyzed (Participants) | 47
  Vomiting-Yes (2011) | 1
  Vomiting-No (2011): number analyzed (Participants) | 47
  Vomiting-No (2011) | 38
  Vomiting-Form not filled (2011): number analyzed (Participants) | 47
  Vomiting-Form not filled (2011) | 0
  Vomiting-Unspecified (2011): number analyzed (Participants) | 47
  Vomiting-Unspecified (2011) | 8
  Diarrhea-Yes (2011): number analyzed (Participants) | 47
  Diarrhea-Yes (2011) | 0
  Diarrhea-No (2011): number analyzed (Participants) | 47
  Diarrhea-No (2011) | 39
  Diarrhea-Form not filled (2011): number analyzed (Participants) | 47
  Diarrhea-Form not filled (2011) | 0
  Diarrhea-Unspecified (2011): number analyzed (Participants) | 47
  Diarrhea-Unspecified (2011) | 8
  Myalgias-Yes (2011): number analyzed (Participants) | 47
  Myalgias-Yes (2011) | 1
  Myalgias-No (2011): number analyzed (Participants) | 47
  Myalgias-No (2011) | 38
  Myalgias-Form not filled (2011): number analyzed (Participants) | 47
  Myalgias-Form not filled (2011) | 0
  Myalgias-Unspecified (2011): number analyzed (Participants) | 47
  Myalgias-Unspecified (2011) | 8
  Nausea-Yes (2011): number analyzed (Participants) | 47
  Nausea-Yes (2011) | 1
  Nausea-No (2011): number analyzed (Participants) | 47
  Nausea-No (2011) | 38
  Nausea-Form not filled (2011): number analyzed (Participants) | 47
  Nausea-Form not filled (2011) | 0
  Nausea-Unspecified (2011): number analyzed (Participants) | 47
  Nausea-Unspecified (2011) | 8
  Headache-Yes (2011): number analyzed (Participants) | 47
  Headache-Yes (2011) | 7
  Headache-No (2011): number analyzed (Participants) | 47
  Headache-No (2011) | 32
  Headache-Form not filled (2011): number analyzed (Participants) | 47
  Headache-Form not filled (2011) | 0
  Headache-Unspecified (2011): number analyzed (Participants) | 47
  Headache-Unspecified (2011) | 8
  Wheezing-Yes (2011): number analyzed (Participants) | 47
  Wheezing-Yes (2011) | 0
  Wheezing-No (2011): number analyzed (Participants) | 47
  Wheezing-No (2011) | 39
  Wheezing-Form not filled (2011): number analyzed (Participants) | 47
  Wheezing-Form not filled (2011) | 0
  Wheezing-Unspecified (2011): number analyzed (Participants) | 47
  Wheezing-Unspecified (2011) | 8
  Apnea-Yes (2011): number analyzed (Participants) | 47
  Apnea-Yes (2011) | 0
  Apnea-No (2011): number analyzed (Participants) | 47
  Apnea-No (2011) | 39
  Apnea-Form not filled (2011): number analyzed (Participants) | 47
  Apnea-Form not filled (2011) | 0
  Apnea-Unspecified (2011): number analyzed (Participants) | 47
  Apnea-Unspecified (2011) | 8
  Tachypnea-Yes (2011): number analyzed (Participants) | 47
  Tachypnea-Yes (2011) | 0
  Tachypnea-No (2011): number analyzed (Participants) | 47
  Tachypnea-No (2011) | 39
  Tachypnea-Form not filled (2011): number analyzed (Participants) | 47
  Tachypnea-Form not filled (2011) | 0
  Tachypnea-Unspecified (2011): number analyzed (Participants) | 47
  Tachypnea-Unspecified (2011) | 8
  Polypnea-Yes (2011): number analyzed (Participants) | 47
  Polypnea-Yes (2011) | 0
  Polypnea-No (2011): number analyzed (Participants) | 47
  Polypnea-No (2011) | 39
  Polypnea-Form not filled (2011): number analyzed (Participants) | 47
  Polypnea-Form not filled (2011) | 0
  Polypnea-Unspecified (2011): number analyzed (Participants) | 47
  Polypnea-Unspecified (2011) | 8
  Arthralgia-Yes (2011): number analyzed (Participants) | 47
  Arthralgia-Yes (2011) | 0
  Arthralgia-No (2011): number analyzed (Participants) | 47
  Arthralgia-No (2011) | 39
  Arthralgia-Form not filled (2011): number analyzed (Participants) | 47
  Arthralgia-Form not filled (2011) | 0
  Arthralgia-Unspecified (2011): number analyzed (Participants) | 47
  Arthralgia-Unspecified (2011) | 8
  Chest Pain-Yes (2011): number analyzed (Participants) | 47
  Chest Pain-Yes (2011) | 0
  Chest Pain-No (2011): number analyzed (Participants) | 47
  Chest Pain-No (2011) | 39
  Chest Pain-Form not filled (2011): number analyzed (Participants) | 47
  Chest Pain-Form not filled (2011) | 0
  Chest Pain-Unspecified (2011): number analyzed (Participants) | 47
  Chest Pain-Unspecified (2011) | 8
  Convulsion-Yes (2011): number analyzed (Participants) | 47
  Convulsion-Yes (2011) | 0
  Convulsion-No (2011): number analyzed (Participants) | 47
  Convulsion-No (2011) | 39
  Convulsion-Form not filled (2011): number analyzed (Participants) | 47
  Convulsion-Form not filled (2011) | 0
  Convulsion-Unspecified (2011): number analyzed (Participants) | 47
  Convulsion-Unspecified (2011) | 8
  Hyporexia-Yes (2011): number analyzed (Participants) | 47
  Hyporexia-Yes (2011) | 0
  Hyporexia-No (2011): number analyzed (Participants) | 47
  Hyporexia-No (2011) | 39
  Hyporexia-Form not filled (2011): number analyzed (Participants) | 47
  Hyporexia-Form not filled (2011) | 0
  Hyporexia-Unspecified (2011): number analyzed (Participants) | 47
  Hyporexia-Unspecified (2011) | 8
  Weakness-Yes (2011): number analyzed (Participants) | 47
  Weakness-Yes (2011) | 4
  Weakness-No (2011): number analyzed (Participants) | 47
  Weakness-No (2011) | 35
  Weakness-Form not filled (2011): number analyzed (Participants) | 47
  Weakness-Form not filled (2011) | 0
  Weakness-Unspecified (2011): number analyzed (Participants) | 47
  Weakness-Unspecified (2011) | 8
  Irritability-Yes (2011): number analyzed (Participants) | 47
  Irritability-Yes (2011) | 0
  Irritability-No (2011): number analyzed (Participants) | 47
  Irritability-No (2011) | 39
  Irritability-Form not filled (2011): number analyzed (Participants) | 47
  Irritability-Form not filled (2011) | 0
  Irritability-Unspecified (2011): number analyzed (Participants) | 47
  Irritability-Unspecified (2011) | 8
  Odynophagia-Yes (2011): number analyzed (Participants) | 47
  Odynophagia-Yes (2011) | 0
  Odynophagia-No (2011): number analyzed (Participants) | 47
  Odynophagia-No (2011) | 39
  Odynophagia-Form not filled (2011): number analyzed (Participants) | 47
  Odynophagia-Form not filled (2011) | 0
  Odynophagia-Unspecified (2011): number analyzed (Participants) | 47
  Odynophagia-Unspecified (2011) | 8
  Abdominal pain-Yes (2011): number analyzed (Participants) | 47
  Abdominal pain-Yes (2011) | 0
  Abdominal pain-No (2011): number analyzed (Participants) | 47
  Abdominal pain-No (2011) | 39
  Abdominal pain-Form not filled (2011): number analyzed (Participants) | 47
  Abdominal pain-Form not filled (2011) | 0
  Abdominal pain-Unspecified (2011): number analyzed (Participants) | 47
  Abdominal pain-Unspecified (2011) | 8
  Conjuntivitis-Yes (2011): number analyzed (Participants) | 47
  Conjuntivitis-Yes (2011) | 0
  Conjuntivitis-No (2011): number analyzed (Participants) | 47
  Conjuntivitis-No (2011) | 39
  Conjuntivitis-Form not filled (2011): number analyzed (Participants) | 47
  Conjuntivitis-Form not filled (2011) | 0
  Conjuntivitis-Unspecified (2011): number analyzed (Participants) | 47
  Conjuntivitis-Unspecified (2011) | 8
  Cyanosis-Yes (2011): number analyzed (Participants) | 47
  Cyanosis-Yes (2011) | 0
  Cyanosis-No (2011): number analyzed (Participants) | 47
  Cyanosis-No (2011) | 39
  Cyanosis-Form not filled (2011): number analyzed (Participants) | 47
  Cyanosis-Form not filled (2011) | 0
  Cyanosis-Unspecified (2011): number analyzed (Participants) | 47
  Cyanosis-Unspecified (2011) | 8
  Chills-Yes (2011): number analyzed (Participants) | 47
  Chills-Yes (2011) | 0
  Chills-No (2011): number analyzed (Participants) | 47
  Chills-No (2011) | 39
  Chills-Form not filled (2011): number analyzed (Participants) | 47
  Chills-Form not filled (2011) | 0
  Chills-Unspecified (2011): number analyzed (Participants) | 47
  Chills-Unspecified (2011) | 8
  Fever-Yes (2012): number analyzed (Participants) | 275
  Fever-Yes (2012) | 252
  Fever-No (2012): number analyzed (Participants) | 275
  Fever-No (2012) | 18
  Fever-Form not filled (2012): number analyzed (Participants) | 275
  Fever-Form not filled (2012) | 0
  Fever-Unspecified (2012): number analyzed (Participants) | 275
  Fever-Unspecified (2012) | 5
  Cough-Yes (2012): number analyzed (Participants) | 275
  Cough-Yes (2012) | 241
  Cough-No (2012): number analyzed (Participants) | 275
  Cough-No (2012) | 26
  Cough-Form not filled (2012): number analyzed (Participants) | 275
  Cough-Form not filled (2012) | 0
  Cough-Unspecified (2012): number analyzed (Participants) | 275
  Cough-Unspecified (2012) | 8
  Sore throat-Yes (2012): number analyzed (Participants) | 275
  Sore throat-Yes (2012) | 120
  Sore throat- No (2012): number analyzed (Participants) | 275
  Sore throat- No (2012) | 146
  Sore throat- Form not filled (2012): number analyzed (Participants) | 275
  Sore throat- Form not filled (2012) | 0
  Sore throat-Unspecified (2012): number analyzed (Participants) | 275
  Sore throat-Unspecified (2012) | 9
  Rhinorrhea-Yes (2012): number analyzed (Participants) | 275
  Rhinorrhea-Yes (2012) | 226
  Rhinorrhea-No (2012): number analyzed (Participants) | 275
  Rhinorrhea-No (2012) | 40
  Rhinorrhea-Form not filled (2012): number analyzed (Participants) | 275
  Rhinorrhea-Form not filled (2012) | 0
  Rhinorrhea-Unspecified (2012): number analyzed (Participants) | 275
  Rhinorrhea-Unspecified (2012) | 9
  Dyspnea-Yes (2012): number analyzed (Participants) | 275
  Dyspnea-Yes (2012) | 27
  Dyspnea-No (2012): number analyzed (Participants) | 275
  Dyspnea-No (2012) | 169
  Dyspnea-Form not filled (2012): number analyzed (Participants) | 275
  Dyspnea-Form not filled (2012) | 0
  Dyspnea-Unspecified (2012): number analyzed (Participants) | 275
  Dyspnea-Unspecified (2012) | 79
  Vomiting-Yes (2012): number analyzed (Participants) | 275
  Vomiting-Yes (2012) | 3
  Vomiting-No (2012): number analyzed (Participants) | 275
  Vomiting-No (2012) | 203
  Vomiting-Form not filled (2012): number analyzed (Participants) | 275
  Vomiting-Form not filled (2012) | 0
  Vomiting-Unspecified (2012): number analyzed (Participants) | 275
  Vomiting-Unspecified (2012) | 69
  Diarrhea-Yes (2012): number analyzed (Participants) | 275
  Diarrhea-Yes (2012) | 5
  Diarrhea-No (2012): number analyzed (Participants) | 275
  Diarrhea-No (2012) | 201
  Diarrhea-Form not filled (2012): number analyzed (Participants) | 275
  Diarrhea-Form not filled (2012) | 0
  Diarrhea-Unspecified (2012): number analyzed (Participants) | 275
  Diarrhea-Unspecified (2012) | 69
  Myalgias-Yes (2012): number analyzed (Participants) | 275
  Myalgias-Yes (2012) | 2
  Myalgias-No (2012): number analyzed (Participants) | 275
  Myalgias-No (2012) | 204
  Myalgias- Form not filled(2012): number analyzed (Participants) | 275
  Myalgias- Form not filled(2012) | 0
  Myalgias-Unspecified (2012): number analyzed (Participants) | 275
  Myalgias-Unspecified (2012) | 69
  Nausea-Yes (2012): number analyzed (Participants) | 275
  Nausea-Yes (2012) | 2
  Nausea-No (2012): number analyzed (Participants) | 275
  Nausea-No (2012) | 204
  Nausea-Form not filled (2012): number analyzed (Participants) | 275
  Nausea-Form not filled (2012) | 0
  Nausea-Unspecified (2012): number analyzed (Participants) | 275
  Nausea-Unspecified (2012) | 69
  Headache-Yes (2012): number analyzed (Participants) | 275
  Headache-Yes (2012) | 33
  Headache-No (2012): number analyzed (Participants) | 275
  Headache-No (2012) | 173
  Headache-Form not filled (2012): number analyzed (Participants) | 275
  Headache-Form not filled (2012) | 0
  Headache-Unspecified (2012): number analyzed (Participants) | 275
  Headache-Unspecified (2012) | 69
  Wheezing-Yes (2012): number analyzed (Participants) | 275
  Wheezing-Yes (2012) | 1
  Wheezing-No (2012): number analyzed (Participants) | 275
  Wheezing-No (2012) | 205
  Wheezing-Form not filled (2012): number analyzed (Participants) | 275
  Wheezing-Form not filled (2012) | 0
  Wheezing-Unspecified (2012): number analyzed (Participants) | 275
  Wheezing-Unspecified (2012) | 69
  Apnea-Yes (2012): number analyzed (Participants) | 275
  Apnea-Yes (2012) | 1
  Apnea-No (2012): number analyzed (Participants) | 275
  Apnea-No (2012) | 205
  Apnea-Form not filled (2012): number analyzed (Participants) | 275
  Apnea-Form not filled (2012) | 0
  Apnea-Unspecified (2012): number analyzed (Participants) | 275
  Apnea-Unspecified (2012) | 69
  Tachypnea-Yes (2012): number analyzed (Participants) | 275
  Tachypnea-Yes (2012) | 0
  Tachypnea-No (2012): number analyzed (Participants) | 275
  Tachypnea-No (2012) | 206
  Tachypnea-Form not filled (2012): number analyzed (Participants) | 275
  Tachypnea-Form not filled (2012) | 0
  Tachypnea-Unspecified (2012): number analyzed (Participants) | 275
  Tachypnea-Unspecified (2012) | 69
  Polypnea-Yes (2012): number analyzed (Participants) | 275
  Polypnea-Yes (2012) | 0
  Polypnea-No (2012): number analyzed (Participants) | 275
  Polypnea-No (2012) | 206
  Polypnea-Form not filled (2012): number analyzed (Participants) | 275
  Polypnea-Form not filled (2012) | 0
  Polypnea-Unspecified (2012): number analyzed (Participants) | 275
  Polypnea-Unspecified (2012) | 69
  Arthralgia-Yes (2012): number analyzed (Participants) | 275
  Arthralgia-Yes (2012) | 0
  Arthralgia-No (2012): number analyzed (Participants) | 275
  Arthralgia-No (2012) | 206
  Arthralgia-Form not filled (2012): number analyzed (Participants) | 275
  Arthralgia-Form not filled (2012) | 0
  Arthralgia-Unspecified (2012): number analyzed (Participants) | 275
  Arthralgia-Unspecified (2012) | 69
  Chest Pain-Yes (2012): number analyzed (Participants) | 275
  Chest Pain-Yes (2012) | 0
  Chest Pain-No (2012): number analyzed (Participants) | 275
  Chest Pain-No (2012) | 206
  Chest Pain-Form not filled (2012): number analyzed (Participants) | 275
  Chest Pain-Form not filled (2012) | 0
  Chest Pain-Unspecified (2012): number analyzed (Participants) | 275
  Chest Pain-Unspecified (2012) | 69
  Convulsion- Yes (2012): number analyzed (Participants) | 275
  Convulsion- Yes (2012) | 0
  Convulsion- No (2012): number analyzed (Participants) | 275
  Convulsion- No (2012) | 206
  Convulsion- Form not filled (2012): number analyzed (Participants) | 275
  Convulsion- Form not filled (2012) | 0
  Convulsion- Unspecified (2012): number analyzed (Participants) | 275
  Convulsion- Unspecified (2012) | 69
  Hyporexia-Yes (2012): number analyzed (Participants) | 275
  Hyporexia-Yes (2012) | 0
  Hyporexia-No (2012): number analyzed (Participants) | 275
  Hyporexia-No (2012) | 206
  Hyporexia-Form not filled (2012): number analyzed (Participants) | 275
  Hyporexia-Form not filled (2012) | 0
  Hyporexia-Unspecified (2012): number analyzed (Participants) | 275
  Hyporexia-Unspecified (2012) | 69
  Weakness-Yes (2012): number analyzed (Participants) | 275
  Weakness-Yes (2012) | 0
  Weakness-No (2012): number analyzed (Participants) | 275
  Weakness-No (2012) | 206
  Weakness-Form not filled (2012): number analyzed (Participants) | 275
  Weakness-Form not filled (2012) | 0
  Weakness-Unspecified (2012): number analyzed (Participants) | 275
  Weakness-Unspecified (2012) | 69
  Irritability-Yes (2012): number analyzed (Participants) | 275
  Irritability-Yes (2012) | 0
  Irritability-No (2012): number analyzed (Participants) | 275
  Irritability-No (2012) | 206
  Irritability-Form not filled (2012): number analyzed (Participants) | 275
  Irritability-Form not filled (2012) | 0
  Irritability-Unspecified (2012): number analyzed (Participants) | 275
  Irritability-Unspecified (2012) | 69
  Odynophagia-Yes (2012): number analyzed (Participants) | 275
  Odynophagia-Yes (2012) | 0
  Odynophagia-No (2012): number analyzed (Participants) | 275
  Odynophagia-No (2012) | 206
  Odynophagia-Form not filled (2012): number analyzed (Participants) | 275
  Odynophagia-Form not filled (2012) | 0
  Odynophagia-Unspecified (2012): number analyzed (Participants) | 275
  Odynophagia-Unspecified (2012) | 69
  Abdominal pain-Yes (2012): number analyzed (Participants) | 275
  Abdominal pain-Yes (2012) | 0
  Abdominal pain-No (2012): number analyzed (Participants) | 275
  Abdominal pain-No (2012) | 206
  Abdominal pain- Form not filled(2012): number analyzed (Participants) | 275
  Abdominal pain- Form not filled(2012) | 0
  Abdominal pain-Unspecified (2012): number analyzed (Participants) | 275
  Abdominal pain-Unspecified (2012) | 69
  Conjuntivitis-Yes (2012): number analyzed (Participants) | 275
  Conjuntivitis-Yes (2012) | 0
  Conjuntivitis-No (2012): number analyzed (Participants) | 275
  Conjuntivitis-No (2012) | 206
  Conjuntivitis-Form not filled (2012): number analyzed (Participants) | 275
  Conjuntivitis-Form not filled (2012) | 0
  Conjuntivitis-Unspecified (2012): number analyzed (Participants) | 275
  Conjuntivitis-Unspecified (2012) | 69
  Cyanosis-Yes (2012): number analyzed (Participants) | 275
  Cyanosis-Yes (2012) | 0
  Cyanosis-No (2012): number analyzed (Participants) | 275
  Cyanosis-No (2012) | 206
  Cyanosis-Form not filled (2012): number analyzed (Participants) | 275
  Cyanosis-Form not filled (2012) | 0
  Cyanosis-Unspecified (2012): number analyzed (Participants) | 275
  Cyanosis-Unspecified (2012) | 69
  Chills-Yes (2012): number analyzed (Participants) | 275
  Chills-Yes (2012) | 0
  Chills-No (2012): number analyzed (Participants) | 275
  Chills-No (2012) | 206
  Chills-Form not filled (2012): number analyzed (Participants) | 275
  Chills-Form not filled (2012) | 0
  Chills-Unspecified (2012): number analyzed (Participants) | 275
  Chills-Unspecified (2012) | 69
  Fever-Yes (2013): number analyzed (Participants) | 190
  Fever-Yes (2013) | 183
  Fever-No (2013): number analyzed (Participants) | 190
  Fever-No (2013) | 5
  Fever-Form not filled (2013): number analyzed (Participants) | 190
  Fever-Form not filled (2013) | 0
  Fever-Unspecified (2013): number analyzed (Participants) | 190
  Fever-Unspecified (2013) | 2
  Cough-Yes (2013): number analyzed (Participants) | 190
  Cough-Yes (2013) | 175
  Cough-No (2013): number analyzed (Participants) | 190
  Cough-No (2013) | 12
  Cough-Form not filled (2013): number analyzed (Participants) | 190
  Cough-Form not filled (2013) | 0
  Cough-Unspecified (2013): number analyzed (Participants) | 190
  Cough-Unspecified (2013) | 3
  Sore throat-Yes (2013): number analyzed (Participants) | 190
  Sore throat-Yes (2013) | 101
  Sore throat-No (2013): number analyzed (Participants) | 190
  Sore throat-No (2013) | 85
  Sore throat-Form not filled (2013): number analyzed (Participants) | 190
  Sore throat-Form not filled (2013) | 0
  Sore throat-Unspecified (2013): number analyzed (Participants) | 190
  Sore throat-Unspecified (2013) | 4
  Rhinorrhea-Yes (2013): number analyzed (Participants) | 190
  Rhinorrhea-Yes (2013) | 168
  Rhinorrhea-No (2013): number analyzed (Participants) | 190
  Rhinorrhea-No (2013) | 18
  Rhinorrhea-Form not filled (2013): number analyzed (Participants) | 190
  Rhinorrhea-Form not filled (2013) | 0
  Rhinorrhea-Unspecified (2013): number analyzed (Participants) | 190
  Rhinorrhea-Unspecified (2013) | 4
  Dyspnea-Yes (2013): number analyzed (Participants) | 190
  Dyspnea-Yes (2013) | 6
  Dyspnea-No (2013): number analyzed (Participants) | 190
  Dyspnea-No (2013) | 125
  Dyspnea-Form not filled (2013): number analyzed (Participants) | 190
  Dyspnea-Form not filled (2013) | 0
  Dyspnea-Unspecified (2013): number analyzed (Participants) | 190
  Dyspnea-Unspecified (2013) | 59
  Vomiting-Yes (2013): number analyzed (Participants) | 190
  Vomiting-Yes (2013) | 3
  Vomiting-No (2013): number analyzed (Participants) | 190
  Vomiting-No (2013) | 142
  Vomiting-Form not filled (2013): number analyzed (Participants) | 190
  Vomiting-Form not filled (2013) | 0
  Vomiting-Unspecified (2013): number analyzed (Participants) | 190
  Vomiting-Unspecified (2013) | 45
  Diarrhea-Yes (2013): number analyzed (Participants) | 190
  Diarrhea-Yes (2013) | 1
  Diarrhea-No (2013): number analyzed (Participants) | 190
  Diarrhea-No (2013) | 144
  Diarrhea-Form not filled (2013): number analyzed (Participants) | 190
  Diarrhea-Form not filled (2013) | 0
  Diarrhea-Unspecified (2013): number analyzed (Participants) | 190
  Diarrhea-Unspecified (2013) | 45
  Myalgias-Yes (2013): number analyzed (Participants) | 190
  Myalgias-Yes (2013) | 5
  Myalgias-No (2013): number analyzed (Participants) | 190
  Myalgias-No (2013) | 140
  Myalgias-Form not filled (2013): number analyzed (Participants) | 190
  Myalgias-Form not filled (2013) | 0
  Myalgias-Unspecified (2013): number analyzed (Participants) | 190
  Myalgias-Unspecified (2013) | 45
  Nausea-Yes (2013): number analyzed (Participants) | 190
  Nausea-Yes (2013) | 2
  Nausea-No (2013): number analyzed (Participants) | 190
  Nausea-No (2013) | 143
  Nausea-Form not filled (2013): number analyzed (Participants) | 190
  Nausea-Form not filled (2013) | 0
  Nausea-Unspecified (2013): number analyzed (Participants) | 190
  Nausea-Unspecified (2013) | 45
  Headache-Yes (2013): number analyzed (Participants) | 190
  Headache-Yes (2013) | 16
  Headache-No (2013): number analyzed (Participants) | 190
  Headache-No (2013) | 129
  Headache-Form not filled (2013): number analyzed (Participants) | 190
  Headache-Form not filled (2013) | 0
  Headache-Unspecified (2013): number analyzed (Participants) | 190
  Headache-Unspecified (2013) | 45
  Wheezing-Yes (2013): number analyzed (Participants) | 190
  Wheezing-Yes (2013) | 0
  Wheezing-No (2013): number analyzed (Participants) | 190
  Wheezing-No (2013) | 145
  Wheezing-Form not filled (2013): number analyzed (Participants) | 190
  Wheezing-Form not filled (2013) | 0
  Wheezing-Unspecified (2013): number analyzed (Participants) | 190
  Wheezing-Unspecified (2013) | 45
  Apnea-Yes (2013): number analyzed (Participants) | 190
  Apnea-Yes (2013) | 0
  Apnea-No (2013): number analyzed (Participants) | 190
  Apnea-No (2013) | 145
  Apnea-Form not filled (2013): number analyzed (Participants) | 190
  Apnea-Form not filled (2013) | 0
  Apnea-Unspecified (2013): number analyzed (Participants) | 190
  Apnea-Unspecified (2013) | 45
  Tachypnea-Yes (2013): number analyzed (Participants) | 190
  Tachypnea-Yes (2013) | 0
  Tachypnea-No (2013): number analyzed (Participants) | 190
  Tachypnea-No (2013) | 145
  Tachypnea-Fom not filled (2013): number analyzed (Participants) | 190
  Tachypnea-Fom not filled (2013) | 0
  Tachypnea-Unspecified (2013): number analyzed (Participants) | 190
  Tachypnea-Unspecified (2013) | 45
  Polypnea-Yes (2013): number analyzed (Participants) | 190
  Polypnea-Yes (2013) | 0
  Polypnea-No (2013): number analyzed (Participants) | 190
  Polypnea-No (2013) | 145
  Polypnea-Form not filled (2013): number analyzed (Participants) | 190
  Polypnea-Form not filled (2013) | 0
  Polypnea-Unspecified (2013): number analyzed (Participants) | 190
  Polypnea-Unspecified (2013) | 45
  Arthralgia-Yes (2013): number analyzed (Participants) | 190
  Arthralgia-Yes (2013) | 0
  Arthralgia-No (2013): number analyzed (Participants) | 190
  Arthralgia-No (2013) | 145
  Arthralgia-Form not filled (2013): number analyzed (Participants) | 190
  Arthralgia-Form not filled (2013) | 0
  Arthralgia-Unspecified (2013): number analyzed (Participants) | 190
  Arthralgia-Unspecified (2013) | 45
  Chest Pain-Yes (2013): number analyzed (Participants) | 190
  Chest Pain-Yes (2013) | 0
  Chest Pain-No (2013): number analyzed (Participants) | 190
  Chest Pain-No (2013) | 145
  Chest Pain-Form not filled (2013): number analyzed (Participants) | 190
  Chest Pain-Form not filled (2013) | 0
  Chest Pain-Unspecified (2013): number analyzed (Participants) | 190
  Chest Pain-Unspecified (2013) | 45
  Convulsion-Yes (2013): number analyzed (Participants) | 190
  Convulsion-Yes (2013) | 0
  Convulsion-No (2013): number analyzed (Participants) | 190
  Convulsion-No (2013) | 145
  Convulsion-Form not filled (2013): number analyzed (Participants) | 190
  Convulsion-Form not filled (2013) | 0
  Convulsion-Unspecified (2013): number analyzed (Participants) | 190
  Convulsion-Unspecified (2013) | 45
  Hyporexia-Yes (2013): number analyzed (Participants) | 190
  Hyporexia-Yes (2013) | 0
  Hyporexia-No (2013): number analyzed (Participants) | 190
  Hyporexia-No (2013) | 145
  Hyporexia-Form not filled (2013): number analyzed (Participants) | 190
  Hyporexia-Form not filled (2013) | 0
  Hyporexia-Unspecified (2013): number analyzed (Participants) | 190
  Hyporexia-Unspecified (2013) | 45
  Weakness-Yes (2013): number analyzed (Participants) | 190
  Weakness-Yes (2013) | 5
  Weakness-No (2013): number analyzed (Participants) | 190
  Weakness-No (2013) | 140
  Weakness-Form not filled (2013): number analyzed (Participants) | 190
  Weakness-Form not filled (2013) | 0
  Weakness-Unspecified (2013): number analyzed (Participants) | 190
  Weakness-Unspecified (2013) | 45
  Irritability-Yes (2013): number analyzed (Participants) | 190
  Irritability-Yes (2013) | 0
  Irritability-No (2013): number analyzed (Participants) | 190
  Irritability-No (2013) | 145
  Irritability-Form not filled (2013): number analyzed (Participants) | 190
  Irritability-Form not filled (2013) | 0
  Irritability-Unspecified (2013): number analyzed (Participants) | 190
  Irritability-Unspecified (2013) | 45
  Odynophagia-Yes (2013): number analyzed (Participants) | 190
  Odynophagia-Yes (2013) | 0
  Odynophagia-No (2013): number analyzed (Participants) | 190
  Odynophagia-No (2013) | 145
  Odynophagia-Form not filled (2013): number analyzed (Participants) | 190
  Odynophagia-Form not filled (2013) | 0
  Odynophagia-Unspecified (2013): number analyzed (Participants) | 190
  Odynophagia-Unspecified (2013) | 45
  Abdominal pain-Yes (2013): number analyzed (Participants) | 190
  Abdominal pain-Yes (2013) | 0
  Abdominal pain-No (2013): number analyzed (Participants) | 190
  Abdominal pain-No (2013) | 145
  Abdominal pain-Form not filled (2013): number analyzed (Participants) | 190
  Abdominal pain-Form not filled (2013) | 0
  Abdominal pain-Unspecified (2013): number analyzed (Participants) | 190
  Abdominal pain-Unspecified (2013) | 45
  Conjuntivitis-Yes (2013): number analyzed (Participants) | 190
  Conjuntivitis-Yes (2013) | 0
  Conjuntivitis-No (2013): number analyzed (Participants) | 190
  Conjuntivitis-No (2013) | 145
  Conjuntivitis-Form not filled (2013): number analyzed (Participants) | 190
  Conjuntivitis-Form not filled (2013) | 0
  Conjuntivitis-Unspecified (2013): number analyzed (Participants) | 190
  Conjuntivitis-Unspecified (2013) | 45
  Cyanosis-Yes (2013): number analyzed (Participants) | 190
  Cyanosis-Yes (2013) | 0
  Cyanosis-No (2013): number analyzed (Participants) | 190
  Cyanosis-No (2013) | 145
  Cyanosis-Form not filled (2013): number analyzed (Participants) | 190
  Cyanosis-Form not filled (2013) | 0
  Cyanosis-Unspecified (2013): number analyzed (Participants) | 190
  Cyanosis-Unspecified (2013) | 45
  Chills-Yes (2013): number analyzed (Participants) | 190
  Chills-Yes (2013) | 2
  Chills-No (2013): number analyzed (Participants) | 190
  Chills-No (2013) | 143
  Chills-Form not filled (2013): number analyzed (Participants) | 190
  Chills-Form not filled (2013) | 0
  Chills-Unspecified (2013): number analyzed (Participants) | 190
  Chills-Unspecified (2013) | 45
  Fever-Yes (2014): number analyzed (Participants) | 140
  Fever-Yes (2014) | 127
  Fever-No (2014): number analyzed (Participants) | 140
  Fever-No (2014) | 10
  Fever-Form not filled (2014): number analyzed (Participants) | 140
  Fever-Form not filled (2014) | 0
  Fever-Unspecified (2014): number analyzed (Participants) | 140
  Fever-Unspecified (2014) | 3
  Cough-Yes (2014): number analyzed (Participants) | 140
  Cough-Yes (2014) | 125
  Cough-No (2014): number analyzed (Participants) | 140
  Cough-No (2014) | 12
  Cough-Form not filled (2014): number analyzed (Participants) | 140
  Cough-Form not filled (2014) | 0
  Cough-Unspecified (2014): number analyzed (Participants) | 140
  Cough-Unspecified (2014) | 3
  Sore throat-Yes (2014): number analyzed (Participants) | 140
  Sore throat-Yes (2014) | 87
  Sore throat-No (2014): number analyzed (Participants) | 140
  Sore throat-No (2014) | 44
  Sore throat-Form not filled (2014): number analyzed (Participants) | 140
  Sore throat-Form not filled (2014) | 0
  Sore throat-Unspecified (2014): number analyzed (Participants) | 140
  Sore throat-Unspecified (2014) | 9
  Rhinorrhea-Yes (2014): number analyzed (Participants) | 140
  Rhinorrhea-Yes (2014) | 101
  Rhinorrhea-No (2014): number analyzed (Participants) | 140
  Rhinorrhea-No (2014) | 34
  Rhinorrhea-Form not filled (2014): number analyzed (Participants) | 140
  Rhinorrhea-Form not filled (2014) | 0
  Rhinorrhea-Unspecified (2014): number analyzed (Participants) | 140
  Rhinorrhea-Unspecified (2014) | 5
  Dyspnea-Yes (2014): number analyzed (Participants) | 140
  Dyspnea-Yes (2014) | 36
  Dyspnea-No (2014): number analyzed (Participants) | 140
  Dyspnea-No (2014) | 76
  Dyspnea-Form not filled (2014): number analyzed (Participants) | 140
  Dyspnea-Form not filled (2014) | 0
  Dyspnea-Unspecified (2014): number analyzed (Participants) | 140
  Dyspnea-Unspecified (2014) | 28
  Vomiting-Yes (2014): number analyzed (Participants) | 140
  Vomiting-Yes (2014) | 0
  Vomiting-No (2014): number analyzed (Participants) | 140
  Vomiting-No (2014) | 117
  Vomiting-Form not filled (2014): number analyzed (Participants) | 140
  Vomiting-Form not filled (2014) | 0
  Vomiting-Unspecified (2014): number analyzed (Participants) | 140
  Vomiting-Unspecified (2014) | 23
  Diarrhea-Yes (2014): number analyzed (Participants) | 140
  Diarrhea-Yes (2014) | 4
  Diarrhea-No (2014): number analyzed (Participants) | 140
  Diarrhea-No (2014) | 113
  Diarrhea-Form not filled (2014): number analyzed (Participants) | 140
  Diarrhea-Form not filled (2014) | 0
  Diarrhea-Unspecified (2014): number analyzed (Participants) | 140
  Diarrhea-Unspecified (2014) | 23
  Myalgias-Yes (2014): number analyzed (Participants) | 140
  Myalgias-Yes (2014) | 3
  Myalgias-No (2014): number analyzed (Participants) | 140
  Myalgias-No (2014) | 114
  Myalgias-Form not filled (2014): number analyzed (Participants) | 140
  Myalgias-Form not filled (2014) | 0
  Myalgias-Unspecified (2014): number analyzed (Participants) | 140
  Myalgias-Unspecified (2014) | 23
  Nausea-Yes (2014): number analyzed (Participants) | 140
  Nausea-Yes (2014) | 1
  Nausea-No (2014): number analyzed (Participants) | 140
  Nausea-No (2014) | 116
  Nausea-Form not filled (2014): number analyzed (Participants) | 140
  Nausea-Form not filled (2014) | 0
  Nausea-Unspecified (2014): number analyzed (Participants) | 140
  Nausea-Unspecified (2014) | 23
  Headache-Yes (2014): number analyzed (Participants) | 140
  Headache-Yes (2014) | 4
  Headache-No (2014): number analyzed (Participants) | 140
  Headache-No (2014) | 113
  Headache-Form not filled (2014): number analyzed (Participants) | 140
  Headache-Form not filled (2014) | 0
  Headache-Unspecified (2014): number analyzed (Participants) | 140
  Headache-Unspecified (2014) | 23
  Wheezing-Yes (2014): number analyzed (Participants) | 140
  Wheezing-Yes (2014) | 0
  Wheezing-No (2014): number analyzed (Participants) | 140
  Wheezing-No (2014) | 117
  Wheezing-Form not filled (2014): number analyzed (Participants) | 140
  Wheezing-Form not filled (2014) | 0
  Wheezing-Unspecified (2014): number analyzed (Participants) | 140
  Wheezing-Unspecified (2014) | 23
  Apnea-Yes (2014): number analyzed (Participants) | 140
  Apnea-Yes (2014) | 0
  Apnea-No (2014): number analyzed (Participants) | 140
  Apnea-No (2014) | 117
  Apnea-Form not filled (2014): number analyzed (Participants) | 140
  Apnea-Form not filled (2014) | 0
  Apnea-Unspecified (2014): number analyzed (Participants) | 140
  Apnea-Unspecified (2014) | 23
  Tachypnea-Yes (2014): number analyzed (Participants) | 140
  Tachypnea-Yes (2014) | 0
  Tachypnea-No (2014): number analyzed (Participants) | 140
  Tachypnea-No (2014) | 117
  Tachypnea-Form not filled (2014): number analyzed (Participants) | 140
  Tachypnea-Form not filled (2014) | 0
  Tachypnea-Unspecified (2014): number analyzed (Participants) | 140
  Tachypnea-Unspecified (2014) | 23
  Polypnea-Yes (2014): number analyzed (Participants) | 140
  Polypnea-Yes (2014) | 0
  Polypnea-No (2014): number analyzed (Participants) | 140
  Polypnea-No (2014) | 117
  Polypnea-Form not filled (2014): number analyzed (Participants) | 140
  Polypnea-Form not filled (2014) | 0
  Polypnea-Unspecified (2014): number analyzed (Participants) | 140
  Polypnea-Unspecified (2014) | 23
  Arthralgia-Yes (2014): number analyzed (Participants) | 140
  Arthralgia-Yes (2014) | 0
  Arthralgia-No (2014): number analyzed (Participants) | 140
  Arthralgia-No (2014) | 117
  Arthralgia-Form not filled (2014): number analyzed (Participants) | 140
  Arthralgia-Form not filled (2014) | 0
  Arthralgia-Unspecified (2014): number analyzed (Participants) | 140
  Arthralgia-Unspecified (2014) | 23
  Chest Pain-Yes (2014): number analyzed (Participants) | 140
  Chest Pain-Yes (2014) | 1
  Chest Pain-No (2014): number analyzed (Participants) | 140
  Chest Pain-No (2014) | 116
  Chest Pain-Form not filled (2014): number analyzed (Participants) | 140
  Chest Pain-Form not filled (2014) | 0
  Chest Pain-Unspecified (2014): number analyzed (Participants) | 140
  Chest Pain-Unspecified (2014) | 23
  Convulsion-Yes (2014): number analyzed (Participants) | 140
  Convulsion-Yes (2014) | 0
  Convulsion-No (2014): number analyzed (Participants) | 140
  Convulsion-No (2014) | 117
  Convulsion-Form not filled (2014): number analyzed (Participants) | 140
  Convulsion-Form not filled (2014) | 0
  Convulsion-Unspecified (2014): number analyzed (Participants) | 140
  Convulsion-Unspecified (2014) | 23
  Hyporexia-Yes (2014): number analyzed (Participants) | 140
  Hyporexia-Yes (2014) | 0
  Hyporexia-No (2014): number analyzed (Participants) | 140
  Hyporexia-No (2014) | 117
  Hyporexia-Form not filled (2014): number analyzed (Participants) | 140
  Hyporexia-Form not filled (2014) | 0
  Hyporexia-Unspecified (2014): number analyzed (Participants) | 140
  Hyporexia-Unspecified (2014) | 23
  Weakness-Yes (2014): number analyzed (Participants) | 140
  Weakness-Yes (2014) | 3
  Weakness-No (2014): number analyzed (Participants) | 140
  Weakness-No (2014) | 114
  Weakness-Form not filled (2014): number analyzed (Participants) | 140
  Weakness-Form not filled (2014) | 0
  Weakness-Unspecified (2014): number analyzed (Participants) | 140
  Weakness-Unspecified (2014) | 23
  Irritability-Yes (2014): number analyzed (Participants) | 140
  Irritability-Yes (2014) | 0
  Irritability-No (2014): number analyzed (Participants) | 140
  Irritability-No (2014) | 117
  Irritability-Form not filled (2014): number analyzed (Participants) | 140
  Irritability-Form not filled (2014) | 0
  Irritability-Unspecified (2014): number analyzed (Participants) | 140
  Irritability-Unspecified (2014) | 23
  Odynophagia-Yes (2014): number analyzed (Participants) | 140
  Odynophagia-Yes (2014) | 0
  Odynophagia-No (2014): number analyzed (Participants) | 140
  Odynophagia-No (2014) | 117
  Odynophagia-Form not filled (2014): number analyzed (Participants) | 140
  Odynophagia-Form not filled (2014) | 0
  Odynophagia-Unspecified (2014): number analyzed (Participants) | 140
  Odynophagia-Unspecified (2014) | 23
  Abdominal pain-Yes (2014): number analyzed (Participants) | 140
  Abdominal pain-Yes (2014) | 0
  Abdominal pain-No (2014): number analyzed (Participants) | 140
  Abdominal pain-No (2014) | 117
  Abdominal pain-Form not filled (2014): number analyzed (Participants) | 140
  Abdominal pain-Form not filled (2014) | 0
  Abdominal pain-Unspecified (2014): number analyzed (Participants) | 140
  Abdominal pain-Unspecified (2014) | 23
  Conjuntivitis-Yes (2014): number analyzed (Participants) | 140
  Conjuntivitis-Yes (2014) | 0
  Conjuntivitis-No (2014): number analyzed (Participants) | 140
  Conjuntivitis-No (2014) | 117
  Conjuntivitis-Form not filled (2014): number analyzed (Participants) | 140
  Conjuntivitis-Form not filled (2014) | 0
  Conjuntivitis-Unspecified (2014): number analyzed (Participants) | 140
  Conjuntivitis-Unspecified (2014) | 23
  Cyanosis-Yes (2014): number analyzed (Participants) | 140
  Cyanosis-Yes (2014) | 0
  Cyanosis-No (2014): number analyzed (Participants) | 140
  Cyanosis-No (2014) | 117
  Cyanosis-Form not filled (2014): number analyzed (Participants) | 140
  Cyanosis-Form not filled (2014) | 0
  Cyanosis-Unspecified (2014): number analyzed (Participants) | 140
  Cyanosis-Unspecified (2014) | 23
  Chills-Yes (2014): number analyzed (Participants) | 140
  Chills-Yes (2014) | 0
  Chills-No (2014): number analyzed (Participants) | 140
  Chills-No (2014) | 117
  Chills-Form not filled (2014): number analyzed (Participants) | 140
  Chills-Form not filled (2014) | 0
  Chills-Unspecified (2014): number analyzed (Participants) | 140
  Chills-Unspecified (2014) | 23
  Fever-Yes (2015): number analyzed (Participants) | 100
  Fever-Yes (2015) | 85
  Fever-No (2015): number analyzed (Participants) | 100
  Fever-No (2015) | 14
  Fever-Form not filled (2015): number analyzed (Participants) | 100
  Fever-Form not filled (2015) | 0
  Fever-Unspecified (2015): number analyzed (Participants) | 100
  Fever-Unspecified (2015) | 1
  Cough-Yes (2015): number analyzed (Participants) | 100
  Cough-Yes (2015) | 88
  Cough-No (2015): number analyzed (Participants) | 100
  Cough-No (2015) | 11
  Cough-Form not filled (2015): number analyzed (Participants) | 100
  Cough-Form not filled (2015) | 0
  Cough-Unspecified (2015): number analyzed (Participants) | 100
  Cough-Unspecified (2015) | 1
  Sore throat-Yes (2015): number analyzed (Participants) | 100
  Sore throat-Yes (2015) | 21
  Sore throat-No (2015): number analyzed (Participants) | 100
  Sore throat-No (2015) | 74
  Sore throat-Form not filled (2015): number analyzed (Participants) | 100
  Sore throat-Form not filled (2015) | 0
  Sore throat-Unspecified (2015): number analyzed (Participants) | 100
  Sore throat-Unspecified (2015) | 5
  Rhinorrhea-Yes (2015): number analyzed (Participants) | 100
  Rhinorrhea-Yes (2015) | 67
  Rhinorrhea-No (2015): number analyzed (Participants) | 100
  Rhinorrhea-No (2015) | 32
  Rhinorrhea-Form not filled (2015): number analyzed (Participants) | 100
  Rhinorrhea-Form not filled (2015) | 0
  Rhinorrhea-Unspecified (2015): number analyzed (Participants) | 100
  Rhinorrhea-Unspecified (2015) | 1
  Dyspnea-Yes (2015): number analyzed (Participants) | 100
  Dyspnea-Yes (2015) | 59
  Dyspnea-No (2015): number analyzed (Participants) | 100
  Dyspnea-No (2015) | 36
  Dyspnea-Form not filled (2015): number analyzed (Participants) | 100
  Dyspnea-Form not filled (2015) | 0
  Dyspnea-Unspecified (2015): number analyzed (Participants) | 100
  Dyspnea-Unspecified (2015) | 5
  Vomiting-Yes (2015): number analyzed (Participants) | 100
  Vomiting-Yes (2015) | 1
  Vomiting-No (2015): number analyzed (Participants) | 100
  Vomiting-No (2015) | 94
  Vomiting-Form not filled (2015): number analyzed (Participants) | 100
  Vomiting-Form not filled (2015) | 0
  Vomiting-Unspecified (2015): number analyzed (Participants) | 100
  Vomiting-Unspecified (2015) | 5
  Diarrhea-Yes (2015): number analyzed (Participants) | 100
  Diarrhea-Yes (2015) | 2
  Diarrhea-No (2015): number analyzed (Participants) | 100
  Diarrhea-No (2015) | 93
  Diarrhea-Form not filled (2015): number analyzed (Participants) | 100
  Diarrhea-Form not filled (2015) | 0
  Diarrhea-Unspecified (2015): number analyzed (Participants) | 100
  Diarrhea-Unspecified (2015) | 5
  Myalgias-Yes (2015): number analyzed (Participants) | 100
  Myalgias-Yes (2015) | 0
  Myalgias-No (2015): number analyzed (Participants) | 100
  Myalgias-No (2015) | 95
  Myalgias-Form not filled (2015): number analyzed (Participants) | 100
  Myalgias-Form not filled (2015) | 0
  Myalgias-Unspecified (2015): number analyzed (Participants) | 100
  Myalgias-Unspecified (2015) | 5
  Nausea-Yes (2015): number analyzed (Participants) | 100
  Nausea-Yes (2015) | 0
  Nausea-No (2015): number analyzed (Participants) | 100
  Nausea-No (2015) | 95
  Nausea-Form not filled (2015): number analyzed (Participants) | 100
  Nausea-Form not filled (2015) | 0
  Nausea-Unspecified (2015): number analyzed (Participants) | 100
  Nausea-Unspecified (2015) | 5
  Headache-Yes (2015): number analyzed (Participants) | 100
  Headache-Yes (2015) | 2
  Headache-No (2015): number analyzed (Participants) | 100
  Headache-No (2015) | 93
  Headache-Form not filled (2015): number analyzed (Participants) | 100
  Headache-Form not filled (2015) | 0
  Headache-Unspecified (2015): number analyzed (Participants) | 100
  Headache-Unspecified (2015) | 5
  Wheezing-Yes (2015): number analyzed (Participants) | 100
  Wheezing-Yes (2015) | 1
  Wheezing-No (2015): number analyzed (Participants) | 100
  Wheezing-No (2015) | 94
  Wheezing-Form not filled (2015): number analyzed (Participants) | 100
  Wheezing-Form not filled (2015) | 0
  Wheezing-Unspecified (2015): number analyzed (Participants) | 100
  Wheezing-Unspecified (2015) | 5
  Apnea-Yes (2015): number analyzed (Participants) | 100
  Apnea-Yes (2015) | 1
  Apnea-No (2015): number analyzed (Participants) | 100
  Apnea-No (2015) | 94
  Apnea-Form not filled (2015): number analyzed (Participants) | 100
  Apnea-Form not filled (2015) | 0
  Apnea-Unspecified (2015): number analyzed (Participants) | 100
  Apnea-Unspecified (2015) | 5
  Tachypnea-Yes (2015): number analyzed (Participants) | 100
  Tachypnea-Yes (2015) | 0
  Tachypnea-No (2015): number analyzed (Participants) | 100
  Tachypnea-No (2015) | 95
  Tachypnea-Form not filled (2015): number analyzed (Participants) | 100
  Tachypnea-Form not filled (2015) | 0
  Tachypnea-Unspecified (2015): number analyzed (Participants) | 100
  Tachypnea-Unspecified (2015) | 5
  Polypnea-Yes (2015): number analyzed (Participants) | 100
  Polypnea-Yes (2015) | 0
  Polypnea-No (2015): number analyzed (Participants) | 100
  Polypnea-No (2015) | 95
  Polypnea-Form not filled (2015): number analyzed (Participants) | 100
  Polypnea-Form not filled (2015) | 0
  Polypnea-Unspecified (2015): number analyzed (Participants) | 100
  Polypnea-Unspecified (2015) | 5
  Arthralgia-Yes (2015): number analyzed (Participants) | 100
  Arthralgia-Yes (2015) | 2
  Arthralgia-No (2015): number analyzed (Participants) | 100
  Arthralgia-No (2015) | 93
  Arthralgia-Form not filled (2015): number analyzed (Participants) | 100
  Arthralgia-Form not filled (2015) | 0
  Arthralgia-Unspecified (2015): number analyzed (Participants) | 100
  Arthralgia-Unspecified (2015) | 5
  Chest Pain-Yes (2015): number analyzed (Participants) | 100
  Chest Pain-Yes (2015) | 1
  Chest Pain-No (2015): number analyzed (Participants) | 100
  Chest Pain-No (2015) | 94
  Chest Pain-Form not filled (2015): number analyzed (Participants) | 100
  Chest Pain-Form not filled (2015) | 0
  Chest Pain-Unspecified (2015): number analyzed (Participants) | 100
  Chest Pain-Unspecified (2015) | 5
  Convulsion-Yes (2015): number analyzed (Participants) | 100
  Convulsion-Yes (2015) | 1
  Convulsion-No (2015): number analyzed (Participants) | 100
  Convulsion-No (2015) | 94
  Convulsion-Form not filled (2015): number analyzed (Participants) | 100
  Convulsion-Form not filled (2015) | 0
  Convulsion-Unspecified (2015): number analyzed (Participants) | 100
  Convulsion-Unspecified (2015) | 5
  Hyporexia-Yes (2015): number analyzed (Participants) | 100
  Hyporexia-Yes (2015) | 0
  Hyporexia-No (2015): number analyzed (Participants) | 100
  Hyporexia-No (2015) | 95
  Hyporexia-Form not filled (2015): number analyzed (Participants) | 100
  Hyporexia-Form not filled (2015) | 0
  Hyporexia-Unspecified (2015): number analyzed (Participants) | 100
  Hyporexia-Unspecified (2015) | 5
  Weakness-Yes (2015): number analyzed (Participants) | 100
  Weakness-Yes (2015) | 0
  Weakness-No (2015): number analyzed (Participants) | 100
  Weakness-No (2015) | 95
  Weakness-Form not filled (2015): number analyzed (Participants) | 100
  Weakness-Form not filled (2015) | 0
  Weakness-Unspecified (2015): number analyzed (Participants) | 100
  Weakness-Unspecified (2015) | 5
  Irritability-Yes (2015): number analyzed (Participants) | 100
  Irritability-Yes (2015) | 0
  Irritability-No (2015): number analyzed (Participants) | 100
  Irritability-No (2015) | 95
  Irritability-Form not filled (2015): number analyzed (Participants) | 100
  Irritability-Form not filled (2015) | 0
  Irritability-Unspecified (2015): number analyzed (Participants) | 100
  Irritability-Unspecified (2015) | 5
  Odynophagia-Yes (2015): number analyzed (Participants) | 100
  Odynophagia-Yes (2015) | 0
  Odynophagia-No (2015): number analyzed (Participants) | 100
  Odynophagia-No (2015) | 95
  Odynophagia-Form not filled (2015): number analyzed (Participants) | 100
  Odynophagia-Form not filled (2015) | 0
  Odynophagia-Unspecified (2015): number analyzed (Participants) | 100
  Odynophagia-Unspecified (2015) | 5
  Abdominal pain-Yes (2015): number analyzed (Participants) | 100
  Abdominal pain-Yes (2015) | 0
  Abdominal pain-No (2015): number analyzed (Participants) | 100
  Abdominal pain-No (2015) | 95
  Abdominal pain-Form not filled (2015): number analyzed (Participants) | 100
  Abdominal pain-Form not filled (2015) | 0
  Abdominal pain-Unspecified (2015): number analyzed (Participants) | 100
  Abdominal pain-Unspecified (2015) | 5
  Conjuntivitis-Yes (2015): number analyzed (Participants) | 100
  Conjuntivitis-Yes (2015) | 0
  Conjuntivitis-No (2015): number analyzed (Participants) | 100
  Conjuntivitis-No (2015) | 95
  Conjuntivitis-Form not filled (2015): number analyzed (Participants) | 100
  Conjuntivitis-Form not filled (2015) | 0
  Conjuntivitis-Unspecified (2015): number analyzed (Participants) | 100
  Conjuntivitis-Unspecified (2015) | 5
  Cyanosis-Yes (2015): number analyzed (Participants) | 100
  Cyanosis-Yes (2015) | 0
  Cyanosis-No (2015): number analyzed (Participants) | 100
  Cyanosis-No (2015) | 95
  Cyanosis-Form not filled (2015): number analyzed (Participants) | 100
  Cyanosis-Form not filled (2015) | 0
  Cyanosis-Unspecified (2015): number analyzed (Participants) | 100
  Cyanosis-Unspecified (2015) | 5
  Chills-Yes (2015): number analyzed (Participants) | 100
  Chills-Yes (2015) | 1
  Chills-No (2015): number analyzed (Participants) | 100
  Chills-No (2015) | 94
  Chills-Form not filled (2015): number analyzed (Participants) | 100
  Chills-Form not filled (2015) | 0
  Chills-Unspecified (2015): number analyzed (Participants) | 100
  Chills-Unspecified (2015) | 5
  Fever-Yes (2016): number analyzed (Participants) | 827
  Fever-Yes (2016) | 686
  Fever-No (2016): number analyzed (Participants) | 827
  Fever-No (2016) | 80
  Fever-Form not filled (2016): number analyzed (Participants) | 827
  Fever-Form not filled (2016) | 24
  Fever-Unspecified (2016): number analyzed (Participants) | 827
  Fever-Unspecified (2016) | 37
  Cough-Yes (2016): number analyzed (Participants) | 827
  Cough-Yes (2016) | 710
  Cough-No (2016): number analyzed (Participants) | 827
  Cough-No (2016) | 49
  Cough-Form not filled (2016): number analyzed (Participants) | 827
  Cough-Form not filled (2016) | 24
  Cough-Unspecified (2016): number analyzed (Participants) | 827
  Cough-Unspecified (2016) | 44
  Sore throat-Yes (2016): number analyzed (Participants) | 827
  Sore throat-Yes (2016) | 351
  Sore throat-No (2016): number analyzed (Participants) | 827
  Sore throat-No (2016) | 356
  Sore throat-Form not filled (2016): number analyzed (Participants) | 827
  Sore throat-Form not filled (2016) | 24
  Sore throat-Unspecified (2016): number analyzed (Participants) | 827
  Sore throat-Unspecified (2016) | 96
  Rhinorrhea-Yes (2016): number analyzed (Participants) | 827
  Rhinorrhea-Yes (2016) | 480
  Rhinorrhea-No (2016): number analyzed (Participants) | 827
  Rhinorrhea-No (2016) | 256
  Rhinorrhea-Form not filled (2016): number analyzed (Participants) | 827
  Rhinorrhea-Form not filled (2016) | 24
  Rhinorrhea-Unspecified (2016): number analyzed (Participants) | 827
  Rhinorrhea-Unspecified (2016) | 67
  Dyspnea-Yes (2016): number analyzed (Participants) | 827
  Dyspnea-Yes (2016) | 372
  Dyspnea-No (2016): number analyzed (Participants) | 827
  Dyspnea-No (2016) | 352
  Dyspnea-Form not filled (2016): number analyzed (Participants) | 827
  Dyspnea-Form not filled (2016) | 24
  Dyspnea-Unspecified (2016): number analyzed (Participants) | 827
  Dyspnea-Unspecified (2016) | 78
  Dyspnea-Missing (2016): number analyzed (Participants) | 827
  Dyspnea-Missing (2016) | 1
  Vomiting-Yes (2016): number analyzed (Participants) | 827
  Vomiting-Yes (2016) | 25
  Vomiting- No (2016): number analyzed (Participants) | 827
  Vomiting- No (2016) | 693
  Vomiting-Form not filled (2016): number analyzed (Participants) | 827
  Vomiting-Form not filled (2016) | 24
  Vomiting-Unspecified (2016): number analyzed (Participants) | 827
  Vomiting-Unspecified (2016) | 85
  Diarrhea-Yes (2016): number analyzed (Participants) | 827
  Diarrhea-Yes (2016) | 25
  Diarrhea-No (2016): number analyzed (Participants) | 827
  Diarrhea-No (2016) | 693
  Diarrhea-Form not filled (2016): number analyzed (Participants) | 827
  Diarrhea-Form not filled (2016) | 24
  Diarrhea-Unspecified (2016): number analyzed (Participants) | 827
  Diarrhea-Unspecified (2016) | 85
  Myalgias-Yes (2016): number analyzed (Participants) | 827
  Myalgias-Yes (2016) | 28
  Myalgias-No (2016): number analyzed (Participants) | 827
  Myalgias-No (2016) | 690
  Myalgias-Form not filled (2016): number analyzed (Participants) | 827
  Myalgias-Form not filled (2016) | 24
  Myalgias-Unspecified (2016): number analyzed (Participants) | 827
  Myalgias-Unspecified (2016) | 85
  Nausea-Yes (2016): number analyzed (Participants) | 827
  Nausea-Yes (2016) | 3
  Nausea-No (2016): number analyzed (Participants) | 827
  Nausea-No (2016) | 715
  Nausea-Form not filled (2016): number analyzed (Participants) | 827
  Nausea-Form not filled (2016) | 24
  Nausea-Unspecified (2016): number analyzed (Participants) | 827
  Nausea-Unspecified (2016) | 85
  Headache-Yes (2016): number analyzed (Participants) | 827
  Headache-Yes (2016) | 45
  Headache-No (2016): number analyzed (Participants) | 827
  Headache-No (2016) | 673
  Headache-Form not filled (2016): number analyzed (Participants) | 827
  Headache-Form not filled (2016) | 24
  Headache-Unspecified (2016): number analyzed (Participants) | 827
  Headache-Unspecified (2016) | 85
  Wheezing-Yes (2016): number analyzed (Participants) | 827
  Wheezing-Yes (2016) | 0
  Wheezing-No (2016): number analyzed (Participants) | 827
  Wheezing-No (2016) | 718
  Wheezing-Form not filled (2016): number analyzed (Participants) | 827
  Wheezing-Form not filled (2016) | 24
  Wheezing-Unspecified (2016): number analyzed (Participants) | 827
  Wheezing-Unspecified (2016) | 85
  Apnea-Yes (2016): number analyzed (Participants) | 827
  Apnea-Yes (2016) | 0
  Apnea-No (2016): number analyzed (Participants) | 827
  Apnea-No (2016) | 718
  Apnea-Form not filled (2016): number analyzed (Participants) | 827
  Apnea-Form not filled (2016) | 24
  Apnea-Unspecified (2016): number analyzed (Participants) | 827
  Apnea-Unspecified (2016) | 85
  Tachypnea-Yes (2016): number analyzed (Participants) | 827
  Tachypnea-Yes (2016) | 2
  Tachypnea-No (2016): number analyzed (Participants) | 827
  Tachypnea-No (2016) | 716
  Tachypnea-Form not filled (2016): number analyzed (Participants) | 827
  Tachypnea-Form not filled (2016) | 24
  Tachypnea-Unspecified (2016): number analyzed (Participants) | 827
  Tachypnea-Unspecified (2016) | 85
  Polypnea-Yes (2016): number analyzed (Participants) | 827
  Polypnea-Yes (2016) | 0
  Polypnea-No (2016): number analyzed (Participants) | 827
  Polypnea-No (2016) | 718
  Polypnea-Form not filled (2016): number analyzed (Participants) | 827
  Polypnea-Form not filled (2016) | 24
  Polypnea-Unspecified (2016): number analyzed (Participants) | 827
  Polypnea-Unspecified (2016) | 85
  Arthralgia-Yes (2016): number analyzed (Participants) | 827
  Arthralgia-Yes (2016) | 7
  Arthralgia-No (2016): number analyzed (Participants) | 827
  Arthralgia-No (2016) | 711
  Arthralgia-Form not filled (2016): number analyzed (Participants) | 827
  Arthralgia-Form not filled (2016) | 24
  Arthralgia-Unspecified (2016): number analyzed (Participants) | 827
  Arthralgia-Unspecified (2016) | 85
  Chest Pain-Yes 2016): number analyzed (Participants) | 827
  Chest Pain-Yes 2016) | 3
  Chest Pain-No (2016): number analyzed (Participants) | 827
  Chest Pain-No (2016) | 715
  Chest Pain-Form not filled (2016): number analyzed (Participants) | 827
  Chest Pain-Form not filled (2016) | 24
  Chest Pain-Unspecified (2016): number analyzed (Participants) | 827
  Chest Pain-Unspecified (2016) | 85
  Convulsion-Yes 2016): number analyzed (Participants) | 827
  Convulsion-Yes 2016) | 5
  Convulsion-No (2016): number analyzed (Participants) | 827
  Convulsion-No (2016) | 713
  Convulsion-Form not filled (2016): number analyzed (Participants) | 827
  Convulsion-Form not filled (2016) | 24
  Convulsion-Unspecified (2016): number analyzed (Participants) | 827
  Convulsion-Unspecified (2016) | 85
  Hyporexia-Yes (2016): number analyzed (Participants) | 827
  Hyporexia-Yes (2016) | 7
  Hyporexia-No (2016): number analyzed (Participants) | 827
  Hyporexia-No (2016) | 711
  Hyporexia-Form not filled (2016): number analyzed (Participants) | 827
  Hyporexia-Form not filled (2016) | 24
  Hyporexia-Unspecified (2016): number analyzed (Participants) | 827
  Hyporexia-Unspecified (2016) | 85
  Weakness-Yes (2016): number analyzed (Participants) | 827
  Weakness-Yes (2016) | 95
  Weakness-No (2016): number analyzed (Participants) | 827
  Weakness-No (2016) | 623
  Weakness-Form not filled (2016): number analyzed (Participants) | 827
  Weakness-Form not filled (2016) | 24
  Weakness-Unspecified (2016): number analyzed (Participants) | 827
  Weakness-Unspecified (2016) | 85
  Irritability-Yes (2016): number analyzed (Participants) | 827
  Irritability-Yes (2016) | 0
  Irritability-No (2016): number analyzed (Participants) | 827
  Irritability-No (2016) | 718
  Irritability-Form not filled (2016): number analyzed (Participants) | 827
  Irritability-Form not filled (2016) | 24
  Irritability-Unspecified (2016): number analyzed (Participants) | 827
  Irritability-Unspecified (2016) | 85
  Odynophagia-Yes (2016): number analyzed (Participants) | 827
  Odynophagia-Yes (2016) | 1
  Odynophagia-No (2016): number analyzed (Participants) | 827
  Odynophagia-No (2016) | 717
  Odynophagia-Form not filled (2016): number analyzed (Participants) | 827
  Odynophagia-Form not filled (2016) | 24
  Odynophagia-Unspecified (2016): number analyzed (Participants) | 827
  Odynophagia-Unspecified (2016) | 85
  Abdominal pain-Yes (2016): number analyzed (Participants) | 827
  Abdominal pain-Yes (2016) | 1
  Abdominal pain-No (2016): number analyzed (Participants) | 827
  Abdominal pain-No (2016) | 717
  Abdominal pain-Form not filled (2016): number analyzed (Participants) | 827
  Abdominal pain-Form not filled (2016) | 24
  Abdominal pain-Unspecified (2016): number analyzed (Participants) | 827
  Abdominal pain-Unspecified (2016) | 85
  Conjuntivitis-Yes (2016): number analyzed (Participants) | 827
  Conjuntivitis-Yes (2016) | 3
  Conjuntivitis-No (2016): number analyzed (Participants) | 827
  Conjuntivitis-No (2016) | 715
  Conjuntivitis-Form not filled (2016): number analyzed (Participants) | 827
  Conjuntivitis-Form not filled (2016) | 24
  Conjuntivitis-Unspecified (2016): number analyzed (Participants) | 827
  Conjuntivitis-Unspecified (2016) | 85
  Cyanosis-Yes (2016): number analyzed (Participants) | 827
  Cyanosis-Yes (2016) | 1
  Cyanosis-No (2016): number analyzed (Participants) | 827
  Cyanosis-No (2016) | 717
  Cyanosis-Form not filled (2016): number analyzed (Participants) | 827
  Cyanosis-Form not filled (2016) | 24
  Cyanosis-Unspecified (2016): number analyzed (Participants) | 827
  Cyanosis-Unspecified (2016) | 85
  Chills-Yes (2016): number analyzed (Participants) | 827
  Chills-Yes (2016) | 7
  Chills-No (2016): number analyzed (Participants) | 827
  Chills-No (2016) | 711
  Chills-Form not filled (2016): number analyzed (Participants) | 827
  Chills-Form not filled (2016) | 24
  Chills-Unspecified (2016): number analyzed (Participants) | 827
  Chills-Unspecified (2016) | 85
  Fever-Yes (2017): number analyzed (Participants) | 260
  Fever-Yes (2017) | 211
  Fever-No (2017): number analyzed (Participants) | 260
  Fever-No (2017) | 42
  Fever-Form not filled (2017): number analyzed (Participants) | 260
  Fever-Form not filled (2017) | 0
  Fever-Unspecified (2017): number analyzed (Participants) | 260
  Fever-Unspecified (2017) | 7
  Cough-Yes (2017): number analyzed (Participants) | 260
  Cough-Yes (2017) | 220
  Cough-No (2017): number analyzed (Participants) | 260
  Cough-No (2017) | 33
  Cough-Form not filled (2017): number analyzed (Participants) | 260
  Cough-Form not filled (2017) | 0
  Cough-Unspecified (2017): number analyzed (Participants) | 260
  Cough-Unspecified (2017) | 7
  Sore throat-Yes (2017): number analyzed (Participants) | 260
  Sore throat-Yes (2017) | 48
  Sore throat-No (2017): number analyzed (Participants) | 260
  Sore throat-No (2017) | 185
  Sore throat-Form not filled (2017): number analyzed (Participants) | 260
  Sore throat-Form not filled (2017) | 0
  Sore throat-Unspecified (2017): number analyzed (Participants) | 260
  Sore throat-Unspecified (2017) | 27
  Rhinorrhea-Yes (2017): number analyzed (Participants) | 260
  Rhinorrhea-Yes (2017) | 189
  Rhinorrhea-No (2017): number analyzed (Participants) | 260
  Rhinorrhea-No (2017) | 56
  Rhinorrhea-Form not filled (2017): number analyzed (Participants) | 260
  Rhinorrhea-Form not filled (2017) | 0
  Rhinorrhea-Unspecified (2017): number analyzed (Participants) | 260
  Rhinorrhea-Unspecified (2017) | 15
  Dyspnea-Yes (2017): number analyzed (Participants) | 260
  Dyspnea-Yes (2017) | 125
  Dyspnea-No (2017): number analyzed (Participants) | 260
  Dyspnea-No (2017) | 101
  Dyspnea-Form not filled (2017): number analyzed (Participants) | 260
  Dyspnea-Form not filled (2017) | 0
  Dyspnea-Unspecified (2017): number analyzed (Participants) | 260
  Dyspnea-Unspecified (2017) | 34
  Vomiting-Yes (2017): number analyzed (Participants) | 260
  Vomiting-Yes (2017) | 7
  Vomiting-No (2017): number analyzed (Participants) | 260
  Vomiting-No (2017) | 219
  Vomiting-Form not filled (2017): number analyzed (Participants) | 260
  Vomiting-Form not filled (2017) | 0
  Vomiting-Unspecified (2017): number analyzed (Participants) | 260
  Vomiting-Unspecified (2017) | 34
  Diarrhea-Yes (2017): number analyzed (Participants) | 260
  Diarrhea-Yes (2017) | 6
  Diarrhea-No (2017): number analyzed (Participants) | 260
  Diarrhea-No (2017) | 220
  Diarrhea-Form not filled (2017): number analyzed (Participants) | 260
  Diarrhea-Form not filled (2017) | 0
  Diarrhea-Unspecified (2017): number analyzed (Participants) | 260
  Diarrhea-Unspecified (2017) | 34
  Myalgias-Yes (2017): number analyzed (Participants) | 260
  Myalgias-Yes (2017) | 4
  Myalgias-No (2017): number analyzed (Participants) | 260
  Myalgias-No (2017) | 222
  Myalgias-Form not filled (2017): number analyzed (Participants) | 260
  Myalgias-Form not filled (2017) | 0
  Myalgias-Unspecified (2017): number analyzed (Participants) | 260
  Myalgias-Unspecified (2017) | 34
  Nausea-Yes (2017): number analyzed (Participants) | 260
  Nausea-Yes (2017) | 0
  Nausea-No (2017): number analyzed (Participants) | 260
  Nausea-No (2017) | 226
  Nausea-Form not filled (2017): number analyzed (Participants) | 260
  Nausea-Form not filled (2017) | 0
  Nausea-Unspecified (2017): number analyzed (Participants) | 260
  Nausea-Unspecified (2017) | 34
  Headache-Yes (2017): number analyzed (Participants) | 260
  Headache-Yes (2017) | 10
  Headache-No (2017): number analyzed (Participants) | 260
  Headache-No (2017) | 216
  Headache-Form not filled (2017): number analyzed (Participants) | 260
  Headache-Form not filled (2017) | 0
  Headache-Unspecified (2017): number analyzed (Participants) | 260
  Headache-Unspecified (2017) | 34
  Wheezing-Yes (2017): number analyzed (Participants) | 260
  Wheezing-Yes (2017) | 1
  Wheezing-No (2017): number analyzed (Participants) | 260
  Wheezing-No (2017) | 225
  Wheezing-Form not filled (2017): number analyzed (Participants) | 260
  Wheezing-Form not filled (2017) | 0
  Wheezing-Unspecified (2017): number analyzed (Participants) | 260
  Wheezing-Unspecified (2017) | 34
  Apnea-Yes (2017): number analyzed (Participants) | 260
  Apnea-Yes (2017) | 0
  Apnea-No (2017): number analyzed (Participants) | 260
  Apnea-No (2017) | 226
  Apnea-Form not filled (2017): number analyzed (Participants) | 260
  Apnea-Form not filled (2017) | 0
  Apnea-Unspecified (2017): number analyzed (Participants) | 260
  Apnea-Unspecified (2017) | 34
  Tachypnea-Yes (2017): number analyzed (Participants) | 260
  Tachypnea-Yes (2017) | 0
  Tachypnea-No (2017): number analyzed (Participants) | 260
  Tachypnea-No (2017) | 226
  Tachypnea-Form not filled (2017): number analyzed (Participants) | 260
  Tachypnea-Form not filled (2017) | 0
  Tachypnea-Unspecified (2017): number analyzed (Participants) | 260
  Tachypnea-Unspecified (2017) | 34
  Polypnea-Yes (2017): number analyzed (Participants) | 260
  Polypnea-Yes (2017) | 0
  Polypnea-No (2017): number analyzed (Participants) | 260
  Polypnea-No (2017) | 226
  Polypnea-Fom not filled (2017): number analyzed (Participants) | 260
  Polypnea-Fom not filled (2017) | 0
  Polypnea-Unspecified (2017): number analyzed (Participants) | 260
  Polypnea-Unspecified (2017) | 34
  Arthralgia-Yes (2017): number analyzed (Participants) | 260
  Arthralgia-Yes (2017) | 2
  Arthralgia-No (2017): number analyzed (Participants) | 260
  Arthralgia-No (2017) | 224
  Arthralgia-Form not filled (2017): number analyzed (Participants) | 260
  Arthralgia-Form not filled (2017) | 0
  Arthralgia-Unspecified (2017): number analyzed (Participants) | 260
  Arthralgia-Unspecified (2017) | 34
  Chest Pain-Yes (2017): number analyzed (Participants) | 260
  Chest Pain-Yes (2017) | 1
  Chest Pain-No (2017): number analyzed (Participants) | 260
  Chest Pain-No (2017) | 225
  Chest Pain-Form not filled (2017): number analyzed (Participants) | 260
  Chest Pain-Form not filled (2017) | 0
  Chest Pain-Unspecified (2017): number analyzed (Participants) | 260
  Chest Pain-Unspecified (2017) | 34
  Convulsion-Yes (2017): number analyzed (Participants) | 260
  Convulsion-Yes (2017) | 2
  Convulsion-No (2017): number analyzed (Participants) | 260
  Convulsion-No (2017) | 224
  Convulsion-Form not filled (2017): number analyzed (Participants) | 260
  Convulsion-Form not filled (2017) | 0
  Convulsion-Unspecified (2017): number analyzed (Participants) | 260
  Convulsion-Unspecified (2017) | 34
  Hyporexia-Yes (2017): number analyzed (Participants) | 260
  Hyporexia-Yes (2017) | 9
  Hyporexia-No (2017): number analyzed (Participants) | 260
  Hyporexia-No (2017) | 217
  Hyporexia-Form not filled (2017): number analyzed (Participants) | 260
  Hyporexia-Form not filled (2017) | 0
  Hyporexia-Unspecified (2017): number analyzed (Participants) | 260
  Hyporexia-Unspecified (2017) | 34
  Weakness-Yes (2017): number analyzed (Participants) | 260
  Weakness-Yes (2017) | 9
  Weakness-No (2017): number analyzed (Participants) | 260
  Weakness-No (2017) | 217
  Weakness-Form not filled (2017): number analyzed (Participants) | 260
  Weakness-Form not filled (2017) | 0
  Weakness-Unspecified (2017): number analyzed (Participants) | 260
  Weakness-Unspecified (2017) | 34
  Irritability-Yes (2017): number analyzed (Participants) | 260
  Irritability-Yes (2017) | 7
  Irritability-No (2017): number analyzed (Participants) | 260
  Irritability-No (2017) | 219
  Irritability-Form not filled (2017): number analyzed (Participants) | 260
  Irritability-Form not filled (2017) | 0
  Irritability-Unspecified (2017): number analyzed (Participants) | 260
  Irritability-Unspecified (2017) | 34
  Odynophagia-Yes (2017): number analyzed (Participants) | 260
  Odynophagia-Yes (2017) | 0
  Odynophagia-No (2017): number analyzed (Participants) | 260
  Odynophagia-No (2017) | 226
  Odynophagia-Form not filled (2017): number analyzed (Participants) | 260
  Odynophagia-Form not filled (2017) | 0
  Odynophagia-Unspecified (2017): number analyzed (Participants) | 260
  Odynophagia-Unspecified (2017) | 34
  Abdominal pain-Yes (2017): number analyzed (Participants) | 260
  Abdominal pain-Yes (2017) | 1
  Abdominal pain-No (2017): number analyzed (Participants) | 260
  Abdominal pain-No (2017) | 225
  Abdominal pain-Form not filled (2017): number analyzed (Participants) | 260
  Abdominal pain-Form not filled (2017) | 0
  Abdominal pain-Unspecified (2017): number analyzed (Participants) | 260
  Abdominal pain-Unspecified (2017) | 34
  Conjuntivitis-Yes (2017): number analyzed (Participants) | 260
  Conjuntivitis-Yes (2017) | 0
  Conjuntivitis-No (2017): number analyzed (Participants) | 260
  Conjuntivitis-No (2017) | 226
  Conjuntivitis-Form not filled (2017): number analyzed (Participants) | 260
  Conjuntivitis-Form not filled (2017) | 0
  Conjuntivitis-Unspecified (2017): number analyzed (Participants) | 260
  Conjuntivitis-Unspecified (2017) | 34
  Cyanosis-Yes (2017): number analyzed (Participants) | 260
  Cyanosis-Yes (2017) | 0
  Cyanosis-No (2017): number analyzed (Participants) | 260
  Cyanosis-No (2017) | 226
  Cyanosis- Form not filled (2017): number analyzed (Participants) | 260
  Cyanosis- Form not filled (2017) | 0
  Cyanosis-Unspecified (2017): number analyzed (Participants) | 260
  Cyanosis-Unspecified (2017) | 34
  Chills-Yes (2017): number analyzed (Participants) | 260
  Chills-Yes (2017) | 0
  Chills-No (2017): number analyzed (Participants) | 260
  Chills-No (2017) | 226
  Chills-Form not filled (2017): number analyzed (Participants) | 260
  Chills-Form not filled (2017) | 0
  Chills-Unspecified (2017): number analyzed (Participants) | 260
  Chills-Unspecified (2017) | 34
  Fever - Yes (Total) | 1585
  Fever - No (Total) | 173
  Fever - Form not filled (Total) | 24
  Fever - Unspecified (Total) | 57
  Cough - Yes (Total) | 1599
  Cough - No (Total) | 147
  Cough - Form not filled (Total) | 24
  Cough - Unspecified (Total) | 69
  Sore throat - Yes (Total) | 754
  Sore throat - No (Total) | 908
  Sore throat - Form not filled (Total) | 24
  Sore throat - Unspecified (Total) | 153
  Rhinorrhea - Yes (Total) | 1272
  Rhinorrhea - No (Total) | 439
  Rhinorrhea - Form not filled (Total) | 24
  Rhinorrhea - Unspecified (Total) | 104
  Dyspnea - Yes (Total) | 629
  Dyspnea - No (Total) | 891
  Dyspnea - Form not filled (Total) | 24
  Dyspnea - Unspecified (Total) | 294
  Dyspnea - Missing (Total) | 1
  Vomiting -Yes (Total) | 40
  Vomiting - No(Total) | 1506
  Vomiting - Form not filled (Total) | 24
  Vomiting - Unspecified (Total) | 269
  Diarrhea - Yes (Total) | 43
  Diarrhea - No (Total) | 1503
  Diarrhea - Form not filled (Total) | 24
  Diarrhea - Unspecified (Total) | 269
  Myalgias - Yes (Total) | 43
  Myalgias - No (Total) | 1503
  Myalgias - Form not filled (Total) | 24
  Myalgias - Unspecified (Total) | 269
  Nausea - Yes (Total) | 9
  Nausea - No (Total) | 1537
  Nausea - Form not filled (Total) | 24
  Nausea - Unspecified (Total) | 269
  Headache - Yes (Total) | 117
  Headache - No (Total) | 1429
  Headache - Form not filled (Total) | 24
  Headache - Unspecified (Total) | 269
  Wheezing - Yes (Total) | 3
  Wheezing - No (Total) | 1543
  Wheezing - Form not filled (Total) | 24
  Wheezing - Unspecified (Total) | 269
  Apnea - Yes (Total) | 2
  Apnea - No (Total) | 1544
  Apnea - Form not filled (Total) | 24
  Apnea - Unspecified (Total) | 269
  Tachypnea - Yes (Total) | 2
  Tachypnea - No (Total) | 1544
  Tachypnea - Form not filled (Total) | 24
  Tachypnea - Unspecified (Total) | 269
  Polypnea - Yes (Total) | 0
  Polypnea - No (Total) | 1546
  Polypnea - Form not filled (Total) | 24
  Polypnea - Unspecified (Total) | 269
  Arthralgia - Yes (Total) | 11
  Arthralgia - No (Total) | 1535
  Arthralgia - Form not filled (Total) | 24
  Arthralgia - Unspecified (Total) | 269
  Chest Pain - Yes (Total) | 6
  Chest Pain - No (Total) | 1540
  Chest Pain - Form not filled (Total) | 24
  Chest Pain - Unspecified (Total) | 269
  Convulsion - Yes (Total) | 8
  Convulsion - No (Total) | 1538
  Convulsion - Form not filled (Total) | 24
  Convulsion - Unspecified (Total) | 269
  Hyporexia- Yes (Total) | 16
  Hyporexia- No (Total) | 1530
  Hyporexia- Form not filled (Total) | 24
  Hyporexia- Unspecified (Total) | 269
  Weakness - Yes (Total) | 116
  Weakness - No (Total) | 1430
  Weakness - Form not filled (Total) | 24
  Weakness - Unspecified (Total) | 269
  Irritability - Yes (Total) | 7
  Irritability - No (Total) | 1539
  Irritability - Form not filled (Total) | 24
  Irritability - Unspecified (Total) | 269
  Odynophagia - Yes (Total) | 1
  Odynophagia - No (Total) | 1545
  Odynophagia - Form not filled (Total) | 24
  Odynophagia - Unspecified (Total) | 269
  Abdominal pain - Yes (Total) | 2
  Abdominal pain - No (Total) | 1544
  Abdominal pain - Form not filled (Total) | 24
  Abdominal pain - Unspecified (Total) | 269
  Conjuntivitis - Yes (Total) | 3
  Conjuntivitis - No (Total) | 1543
  Conjuntivitis - Form not filled (Total) | 24
  Conjuntivitis - Unspecified (Total) | 269
  Cyanosis - Yes (Total) | 1
  Cyanosis - No (Total) | 1545
  Cyanosis - Form not filled (Total) | 24
  Cyanosis - Unspecified (Total) | 269
  Chills - Yes (Total) | 10
  Chills - No (Total) | 1536
  Chills - Form not filled (Total) | 24
  Chills - Unspecified (Total) | 269

5. Secondary Outcome: Number of Cases With Laboratory Confirmed Diagnosis Seasonal Influenza A and/or B Who Experienced Outcomes (Complications)
Description: The outcomes were categorized as follows: Outpatient, Hospitalised, Dead or Unspecified (i.e. missing data on the epidemiology surveillance form). Note that one specimen sample was positive for both influenza A and B so the number started still remains 1839.
Time Frame: From January 2011 to December 2017
Population: The analysis was performed on the Total Cohort which included specimen samples diagnosed with seasonal influenza A and/or B, reported in the ICGES database of Panama, from January 2011 to December 2017.
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza Virus Positive Group
Number analyzed (Participants) | 1839
Participants
  Outpatient (2011): number analyzed (Participants) | 47
  Outpatient (2011) | 37
  Hospitalised (2011): number analyzed (Participants) | 47
  Hospitalised (2011) | 10
  Dead (2011): number analyzed (Participants) | 47
  Dead (2011) | 0
  Unspecified (2011): number analyzed (Participants) | 47
  Unspecified (2011) | 0
  Outpatient (2012): number analyzed (Participants) | 275
  Outpatient (2012) | 132
  Hospitalised (2012): number analyzed (Participants) | 275
  Hospitalised (2012) | 79
  Dead (2012): number analyzed (Participants) | 275
  Dead (2012) | 0
  Unspecified (2012): number analyzed (Participants) | 275
  Unspecified (2012) | 64
  Outpatient (2013): number analyzed (Participants) | 190
  Outpatient (2013) | 119
  Hospitalised (2013): number analyzed (Participants) | 190
  Hospitalised (2013) | 59
  Dead (2013): number analyzed (Participants) | 190
  Dead (2013) | 0
  Unspecified (2013): number analyzed (Participants) | 190
  Unspecified (2013) | 12
  Outpatient (2014): number analyzed (Participants) | 140
  Outpatient (2014) | 90
  Hospitalised (2014): number analyzed (Participants) | 140
  Hospitalised (2014) | 50
  Dead (2014): number analyzed (Participants) | 140
  Dead (2014) | 0
  Unspecified (2014): number analyzed (Participants) | 140
  Unspecified (2014) | 0
  Outpatient (2015): number analyzed (Participants) | 100
  Outpatient (2015) | 24
  Hospitalised (2015): number analyzed (Participants) | 100
  Hospitalised (2015) | 76
  Dead (2015): number analyzed (Participants) | 100
  Dead (2015) | 0
  Unspecified (2015): number analyzed (Participants) | 100
  Unspecified (2015) | 0
  Outpatient (2016): number analyzed (Participants) | 827
  Outpatient (2016) | 338
  Hospitalised (2016): number analyzed (Participants) | 827
  Hospitalised (2016) | 465
  Dead (2016): number analyzed (Participants) | 827
  Dead (2016) | 10
  Unspecified (2016): number analyzed (Participants) | 827
  Unspecified (2016) | 14
  Outpatient (2017): number analyzed (Participants) | 260
  Outpatient (2017) | 66
  Hospitalised (2017): number analyzed (Participants) | 260
  Hospitalised (2017) | 192
  Dead (2017): number analyzed (Participants) | 260
  Dead (2017) | 1
  Unspecified (2017): number analyzed (Participants) | 260
  Unspecified (2017) | 1
  Outpatient (Total) | 806
  Hospitalised (Total) | 931
  Dead (Total) | 11
  Unspecified (Total) | 91

6. Secondary Outcome: Number of Seasonal Influenza A and /or B Cases by Southern Hemisphere, Within Different Seasons From 2011 to 2017
Description: The cases were stratified by influenza type and Southern hemisphere Influenza seasonal period (May-October of each year 2011-2017). Note that one specimen sample was positive for both influenza A and B so the number started still remains 1839.
Time Frame: Within the Southern hemisphere influenza seasons (May to October of each year 2011-2017)
Population: The analysis was performed on the Total Cohort which included all specimen samples diagnosed with seasonal influenza A and/or B, reported in the ICGES database of Panama, within the Southern hemisphere influenza seasons (May to October of each year 2011-2017).
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza Virus Positive Group
Number analyzed (Participants) | 1580
Participants
  Influenza A (May-Oct 2011): number analyzed (Participants) | 41
  Influenza A (May-Oct 2011) | 41
  Influenza B (May-Oct 2011): number analyzed (Participants) | 41
  Influenza B (May-Oct 2011) | 0
  Influenza A (May-Oct 2012): number analyzed (Participants) | 264
  Influenza A (May-Oct 2012) | 93
  Influenza B (May-Oct 2012): number analyzed (Participants) | 264
  Influenza B (May-Oct 2012) | 172
  Influenza A (May-Oct 2013): number analyzed (Participants) | 177
  Influenza A (May-Oct 2013) | 177
  Influenza B (May-Oct 2013): number analyzed (Participants) | 177
  Influenza B (May-Oct 2013) | 0
  Influenza A (May-Oct 2014): number analyzed (Participants) | 104
  Influenza A (May-Oct 2014) | 50
  Influenza B (May-Oct 2014): number analyzed (Participants) | 104
  Influenza B (May-Oct 2014) | 54
  Influenza A (May-Oct 2015): number analyzed (Participants) | 74
  Influenza A (May-Oct 2015) | 74
  Influenza B (May-Oct 2015): number analyzed (Participants) | 74
  Influenza B (May-Oct 2015) | 0
  Influenza A (May-Oct 2016): number analyzed (Participants) | 698
  Influenza A (May-Oct 2016) | 698
  Influenza B (May-Oct 2016): number analyzed (Participants) | 698
  Influenza B (May-Oct 2016) | 0
  Influenza A (May-Oct 2017): number analyzed (Participants) | 222
  Influenza A (May-Oct 2017) | 91
  Influenza B (May-Oct 2017): number analyzed (Participants) | 222
  Influenza B (May-Oct 2017) | 131
  Influenza A (total for all seasons 2011-2017) | 1224
  Influenza B (total for all seasons (2011-2017) | 357

7. Secondary Outcome: Number of Seasonal Influenza A and /or B Cases by Region, Within Study Period From 2011 to 2017
Description: The cases were stratified by region. Regions were classified as follows: West, Central, Panama, Northeast, Unspecified (= region unknown). Note that one specimen sample was positive for both influenza A and B so the number started still remains 1839.
Time Frame: From January 2011 to December 2017
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza Virus Positive Group
Number analyzed (Participants) | 1839
Participants
  Influenza A (West): number analyzed (Participants) | 427
  Influenza A (West) | 345
  Influenza B (West): number analyzed (Participants) | 427
  Influenza B (West) | 82
  Influenza A (Central): number analyzed (Participants) | 308
  Influenza A (Central) | 244
  Influenza B (Central): number analyzed (Participants) | 308
  Influenza B (Central) | 64
  Influenza A (Panama): number analyzed (Participants) | 1006
  Influenza A (Panama) | 805
  Influenza B (Panama): number analyzed (Participants) | 1006
  Influenza B (Panama) | 201
  Influenza A (Northeast): number analyzed (Participants) | 59
  Influenza A (Northeast) | 48
  Influenza B (Northeast): number analyzed (Participants) | 59
  Influenza B (Northeast) | 12
  Influenza A (Unspecified): number analyzed (Participants) | 39
  Influenza A (Unspecified) | 22
  Influenza B (Unspecified): number analyzed (Participants) | 39
  Influenza B (Unspecified) | 17
  Influenza A (Total) | 1464
  Influenza B (Total) | 376

8. Secondary Outcome: Number of Influenza Cases Caused by B- Strain and Presented by B-lineage and by Region Among All Influenza Cases A and/or B
Description: The cases were stratified by lineage (Victoria and Yamagata) and region. Regions were classified as follows: West, Central, Panama, Northeast, Unspecified (= region unknown). Note that one specimen sample was positive for both influenza A and B so the number started still remains 1839.
Time Frame: From January 2011 to December 2017
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza Virus Positive Group
Number analyzed (Participants) | 1839
Participants
  Victoria (West): number analyzed (Participants) | 427
  Victoria (West) | 61
  Yamagata (West): number analyzed (Participants) | 427
  Yamagata (West) | 21
  Victoria (Central): number analyzed (Participants) | 308
  Victoria (Central) | 48
  Yamagata (Central): number analyzed (Participants) | 308
  Yamagata (Central) | 16
  Victoria (Panama): number analyzed (Participants) | 1006
  Victoria (Panama) | 138
  Yamagata (Panama): number analyzed (Participants) | 1006
  Yamagata (Panama) | 63
  Victoria (Northeast): number analyzed (Participants) | 59
  Victoria (Northeast) | 5
  Yamagata (Northeast): number analyzed (Participants) | 59
  Yamagata (Northeast) | 7
  Victoria (Unspecified): number analyzed (Participants) | 39
  Victoria (Unspecified) | 17
  Yamagata (Unspecified): number analyzed (Participants) | 39
  Yamagata (Unspecified) | 0
  Victoria (Total) | 269
  Yamagata (Total) | 107

9. Secondary Outcome: Number of Circulating Influenza B Lineage Positive Specimens Mismatch With the B-strain Vaccine Recommendation, Among the Number of Influenza B Positive Specimens, by Influenza Seasons
Description: Comparison of characteristics of the influenza B-infection Victoria (V) or Yamagata (Y) as observed in the database and the B-strain included in the trivalent influenza vaccine expressed as the number of cases with B-lineage-level mismatch between trivalent seasonal influenza vaccines and circulating viruses observed during the study period. Categories are defined as follows: e.g. for the first category:"V.(B/Brisbane/60/2008)vsVictoria-May-Oct 2011" corresponds to Southern hemisphere influenza season of "May-Oct 2011" with vaccine recommendation: "Victoria (B/Brisbane/60/2008-like virus)" compared to circulating Influenza B lineages "Victoria". Note that one specimen sample was positive for both influenza A and B so the number started still remains 1839.
Time Frame: Within the Southern hemisphere influenza seasons (May to October of each year 2011-2017)
Population: The analysis was performed on the specimen samples, among the Total Cohort, diagnosed with seasonal influenza B, reported in the ICGES database of Panama, within the Southern hemisphere influenza seasons (May to October of each year 2011-2017).
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza Virus Positive Group
Number analyzed (Participants) | 357
Participants
  V.(B/Brisbane/60/2008)vsVictoria-May-Oct 2011: number analyzed (Participants) | 0
  V.(B/Brisbane/60/2008)vsYamagata-May-Oct 2011: number analyzed (Participants) | 0
  V.(B/Brisbane/60/2008)vsVictoria-May-Oct 2012: number analyzed (Participants) | 172
  V.(B/Brisbane/60/2008)vsVictoria-May-Oct 2012 | 172
  V.(B/Brisbane/60/2008)vsYamagata-May-Oct 2012: number analyzed (Participants) | 172
  V.(B/Brisbane/60/2008)vsYamagata-May-Oct 2012 | 0
  Y.(B/Wisconsin/1/2010)vsVictoria-May-Oct 2013: number analyzed (Participants) | 0
  Y.(B/Wisconsin/1/2010)vsYamagata-May-Oct 2013: number analyzed (Participants) | 0
  Y.(B/Massachusetts/2/2012)vsVictoria-May-Oct 2014: number analyzed (Participants) | 54
  Y.(B/Massachusetts/2/2012)vsVictoria-May-Oct 2014 | 0
  Y.(B/Massachusetts/2/2012)vsYamagata-May-Oct 2014: number analyzed (Participants) | 54
  Y.(B/Massachusetts/2/2012)vsYamagata-May-Oct 2014 | 54
  Y.(B/Phuket/3073/2013)vsVictoria-May-Oct 2015: number analyzed (Participants) | 0
  Y.(B/Phuket/3073/2013)vsYamagata-May-Oct 2015: number analyzed (Participants) | 0
  V.(B/Brisbane/60/2008)vsVictoria-May-Oct 2016: number analyzed (Participants) | 0
  V.(B/Brisbane/60/2008)vsYamagata-May-Oct 2016: number analyzed (Participants) | 0
  V.(B/Brisbane/60/2008)vsVictoria-May-Oct 2017: number analyzed (Participants) | 131
  V.(B/Brisbane/60/2008)vsVictoria-May-Oct 2017 | 80
  V.(B/Brisbane/60/2008)vsYamagata-May-Oct 2017: number analyzed (Participants) | 131
  V.(B/Brisbane/60/2008)vsYamagata-May-Oct 2017 | 51

ADVERSE EVENTS:
Time Frame: No safety data have been collected in the study.
Description: There was no subject enrolment in the study. The study encompassed subject specimen samples reported in the ICGES database of Panama.
Arm/Group | Influenza Virus Positive Group
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-03-29): https://cdn.clinicaltrials.gov/large-docs/46/NCT02885246/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-20): https://cdn.clinicaltrials.gov/large-docs/46/NCT02885246/SAP_001.pdf